CLINICAL TRIAL: NCT03020745
Title: A Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Dose and Multiple Doses of GSK3389404 in Chronic Hepatitis B Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of GSK3389404 in Chronic Hepatitis B (CHB) Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 205670
Record Dates: First submitted 2016-12-05; First posted 2017-01-13 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Hepatitis B
Keywords: Pharmacokinetics; Safety; Pharmacodynamics; Efficacy; Chronic Hepatitis B; GSK3389404
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1, Cohort A : GSK3389404 30 mg SC or Placebo (Experimental): Enrolled subjects (HBeAg-positive and/or HBeAg negative) will receive single SC injection of GSK3389404 30 mg or matching placebo
  Interventions: Drug: GSK3389404; Drug: Placebo
- Part 1, Cohort B: GSK3389404 60 mg SC or Placebo (Experimental): Enrolled subjects (HBeAg-positive and/or HBeAg negative) will receive single SC injection of GSK3389404 60 mg or matching placebo
  Interventions: Drug: GSK3389404; Drug: Placebo
- Part 1, Cohort C: GSK3389404 120 mg SC or Placebo (Experimental): Enrolled subjects (HBeAg-positive and/or HBeAg negative) will receive single SC injection of GSK3389404 120 mg or matching placebo
  Interventions: Drug: GSK3389404; Drug: Placebo
- Part 1, Cohort C1 (optional): GSK3389404 120 mg SC or Placebo (Experimental): Enrolled subjects (HBeAg-positive and/or HBeAg negative) will receive single SC injection of GSK3389404 120 mg or matching placebo
  Interventions: Drug: GSK3389404; Drug: Placebo
- Part 1, Cohort D: GSK3389404 </= 240 mg SC or Placebo (Experimental): Enrolled subjects (HBeAg-positive and/or HBeAg negative) will receive single SC injection of GSK3389404 <= 240 mg or matching placebo
  Interventions: Drug: GSK3389404; Drug: Placebo
- Part 2: GSK3389404 or placebo SC (Experimental): Enrolled subjects will receive different parallel dose level and regimens of GSK3389404 or placebo SC at dose determined in part 1. The treatments for Part 2 are 60 mg GSK3389404 weekly, 120 mg bi-weekly GSK3389404, 120 mg GSK3389404 weekly or placebo.
  Interventions: Drug: GSK3389404; Drug: Placebo

INTERVENTIONS:
Drug: GSK3389404 — GSK3389404 is available as Clear colorless to slightly yellow solution for injection.
Drug: Placebo — Placebo is available as a Clear colorless solution.

SUMMARY:
GSK3389404 is being developed for the treatment of CHB virus infection. The development goal for GSK3389404 is the establishment of a finite duration treatment that results in sustained suppression of hepatitis B virus (HBV) replication and viral antigen production after cessation of all treatments for CHB due to the restoration of a functional immune response in the absence of high antigen levels. This study is a multicenter, randomized double-Blind (sponsor un-blinded in Part 1), Placebo-controlled Study which will evaluate the safety, tolerability, PK, and PD profile of GSK3389404 in subjects with CHB and aim to establish proof-of-mechanism. The study will be conducted in two parts. Part 1 plans to enroll subjects primarily from the Asia-pacific region, including Japan and will be conducted as a single ascending dose (SAD) study with 5 planned cohorts ranging from 30 milligram (mg) to a maximum of 240 mg GSK3389404. Within each cohort, subjects will be randomized to receive either GSK3389404 or placebo in a 3:1 ratio. Cohorts A, B, C, C1, and D will be conducted in a sequential fashion; Cohort C1 is an optional cohort and may be dosed after Cohort C or in parallel with Cohort D. Part 2 will be conducted as a multiple-dose, dose-ranging study. Subjects will be randomized to different parallel dose levels and regimens or placebo. The dose levels of Part 2 will be selected after a review of Part 1 safety, Pharmacokinetic (PK) and Pharmacodynamic (PD) data. The treatments selected are 60 mg GSK3389404 weekly, 120 mg GSK3389404 bi-weekly, 120 mg GSK3389404 weekly or placebo. An optional Japanese part-2 sub-study is planned. The total study duration for part 1 including screening, treatment, and post-treatment follow-up, will not be expected to exceed 13 weeks for each subject and for part 2, including screening, treatment and post-treatment follow-up, will not be expected to exceed 65 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand and is capable of giving written informed consent, is willing to comply with protocol requirements, instructions and protocol-stated restrictions, and is likely to complete the study as planned.
* Between 18 and 70 years of age, inclusive, at the time of signing the informed consent form.
* A body mass index (BMI) between 18 to 30 kilogram (Kg)/meter (m^2), inclusive.
* Male or female if they satisfy the following: All females must meet the following criteria: Non-pregnant (as confirmed by a negative serum Human Chorionic Gonadotropin [hCG] test); AND Non-lactating at screening and prior to dosing; AND For Part 2, females of reproductive potential (FRP) must agree to follow (or confirm that they have and are currently following) one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP from at least 28 days prior to the first dose of study treatment until Follow-up visit Day 169 in conjunction with partner's use of male condom. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. For females of non-reproductive potential at least one of the following conditions must apply: Premenopausal females without reproductive potential defined by Documented salpingectomy, Hysterectomy or Documented bilateral oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea; A blood sample for simultaneous Follicle-Stimulating Hormone (FSH) and estradiol levels may be collected at the discretion of the investigator or site to confirm non-reproductive potential; Male subjects with a female partner of child-bearing potential must agree to meet one of the contraception requirements from the time of first dose of study treatment until Follow-up visit Day 169; Vasectomy; Male condom plus partner's use of one of the contraceptive options below that meets the Standard Operating Procedure (SOP) effectiveness criteria including a <1 percent rate of failure per year, as stated in the product label: Contraceptive subdermal implant, Intrauterine device or intrauterine system, Combined estrogen and progestogen oral contraceptive, Injectable progestogen, Contraceptive vaginal ring, or Percutaneous contraceptive patches. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. Male subjects must refrain from donating sperm from the time of first dose of study treatment until Follow-up visit Day 169.
* Documented chronic HBV infection >=6 months prior to screening.
* Subjects with HBV treatment history as follows: Part 1: Treatment naive or have had prior treatment with interferon (pegylated or non pegylated) that must have ended at least 6 months prior to the Baseline visit (Day 1 pre-dose) and/or nucleos(t)ide analogue therapy that must have ended at least 6 months prior to the Baseline visit or currently receiving stable nucleos(t)ide analogue therapy, defined as no changes to their nucleos(t)ide regimen from at least 6 months prior to screening and with no planned changes to the stable regimen over the duration of the study. Part 2: Subjects with CHB receiving stable nucleos(t)ide analogue therapy, defined as no changes to their nucleos(t)ide regimen from at least 6 months prior to screening and with no planned changes to the stable regimen over the duration of the study. Subjects with prior treatment with interferon (pegylated or non-pegylated) must have ended treatment at least 6 months prior to the Baseline visit (Day 1 pre-dose).
* Plasma or serum HBV DNA concentration: treatment naïve subjects or subjects not currently receiving treatment, there is no minimum HBV DNA requirement; Subjects who are receiving stable nucleos(t)ide analogue therapy must be adequately suppressed, defined as plasma or serum HBV DNA <lower limit of quantification (LLOQ)
* Plasma or serum HBsAg concentration >50 IU/mL.
* Alanine aminotransferase (ALT) concentration: ALT < 5 X Upper Limit of Normal (ULN) for treatment naïve subjects and for subjects who are not currently receiving treatment. ALT <=2 times ULN for subjects who are receiving stable nucleos(t)ide analogue therapy.

Exclusion Criteria:

* Medical history: History of or active diagnosis of moderate to severe liver disease other than CHB, such as autoimmune hepatitis, non alcoholic steatohepatitis, hemochromatosis, or liver failure. History or other clinical evidence of significant or unstable cardiac disease (e.g., prolonged QT syndrome [torsade de pointes], angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease and/or clinically significant ECG abnormalities). Uncontrolled or history of difficult to control hypertension. History of, or active diagnosis of, primary or secondary renal disease (e.g., renal disease secondary to diabetes, hypertension, vascular disease, etc.). History of extrahepatic disorders possibly related to HBV immune complexes (e.g., glomerulonephritis and polyarteritis nodosa). History of bleeding diathesis or coagulopathy. History of or suspected presence of vasculitis. History of Gilbert's Syndrome. History of malignancy within the past 5 years with the exception of specific cancers that are cured by surgical resection (e.g., skin cancer), subjects under evaluation for possible malignancy are not eligible.
* History of/sensitivity to GSK3389404 or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Confirmed or suspected hepatocellular carcinoma (HCC) as evidenced by: Alpha-fetoprotein concentration >=200 nanogram (ng)/mL. If the screening alpha-fetoprotein concentration is >=50 ng/mL and <200 ng/mL, the absence of liver mass must be documented by imaging within 6 months before randomization.
* Liver cirrhosis or evidence of cirrhosis as determined by any of the following: Positive liver biopsy (i.e., Metavir Score F4) within 12 months of screening. Fibroscan >12 kilopascals (kPa) within 12 months of screening. AST-Platelet Index (APRI) >2 and FibroSure result >0.7 within 12 months of screening and Investigator judgment. For subjects without a test for cirrhosis in the above timeframes, APRI and FibroSure should be performed during the screening period to rule out cirrhosis.
* Hepatitis C Virus (HCV) co-infection.
* Human Immunodeficiency Virus (HIV) co-infection.
* Hepatitis D Virus (HDV) co-infection.
* Laboratory results as follows: Total bilirubin concentration >1.25 X ULN. Serum albumin concentration <3.5 grams (g)/deciliter (dL). International normalized ratio (INR) >1.25. Platelet count <140 X 10^9/L. Serum creatinine concentration greater than the ULN. Glomerular Filtration Rate (GFR) <90 mL/min as calculated by the Chronic Kidney Disease Epidemiologic Collaboration (CKD-EPI) formula. Subjects with GFR <90 mL/min but >= 60 mL/min may be considered after consultation with the GlaxoSmithKline medical monitor. Urine Albumin to Creatinine Ratio (ACR)>=0.03 mg/mg (or >=30 mg/g). In the event of an ACR above this threshold, eligibility may be confirmed by a second measurement in cases where subjects have low urine albumin and low urine creatinine levels resulting in a urine ACR calculation >=0.03 mg/mg (or >=30 mg/g), the investigator should confirm that subject does not have a history of diabetes, hypertension or other risk factors that may affect renal function and discuss with the PPD or GSK medical monitor, or designee.
* Positive test for blood in urine. In the event of a positive test, the test may be repeated once, and if repeat is negative or if urine microscopy reveals <5 RBC per High-Power Field (HPF), the subject is considered eligible.
* Fridericia's QT correction formula (QTcF) >=450 milliseconds (msec) (single ECG at screening shows QTcF >=450 msec, a mean of triplicate measurements should be used to confirm that subject meets exclusion criterion).
* Currently taking, or took within 3 months of screening, any immunosuppressing drugs (e.g., prednisone), other than a short course of therapy (<=2 weeks) or topical/inhaled steroid use.
* Current alcohol use as judged by investigator to potentially interfere with participant compliance.
* A positive pre-study treatment screen and an unwillingness to refrain from use of illicit drugs (or substances with abuse potential) and adhere to other protocol-stated restrictions while participating in the study [The screen refers to illicit drugs and substances with abuse potential. Medications that are used by the subject as directed, whether over-the-counter or through prescription, are acceptable and would not meet the exclusion criteria]. .
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 5 half-lives (if known) or twice the duration (if known) of the biological effect of the study treatment (whichever is longer) or 90 days (if half-life or duration is unknown).
* Prior treatment with any non-GSK oligonucleotide or small interfering ribonucleic acid (RNA) (siRNA) within 12 months prior to the first dosing day or prior treatment with GSK oligonucleotide within 3 months prior to the first dosing day.
* Pregnant or lactating females at screening and prior to dosing.
* For Part 1, females of reproductive potential.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- China (3):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
- GSK Investigational Site, Pokfulam, Hong Kong
- Japan (5):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaidou
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Tokyo
- Philippines (2):
  - GSK Investigational Site, Cebu
  - GSK Investigational Site, Makati City
- GSK Investigational Site, Singapore, Singapore
- South Korea (4):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request Site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Han K, Theodore D, McMullen G, Swayze E, McCaleb M, Billioud G, Wieland S, Hood S, Paff M, Bennett CF, Kwoh TJ. Preclinical and Phase 1 Assessment of Antisense Oligonucleotide Bepirovirsen in Hepatitis B Virus-Transgenic Mice and Healthy Human Volunteers: Support for Clinical Dose Selection and Evaluation of Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses. Clin Pharmacol Drug Dev. 2022 Oct;11(10):1191-1202. doi: 10.1002/cpdd.1154. Epub 2022 Aug 16. PMID 35971951
- [Derived] Yuen MF, Heo J, Kumada H, Suzuki F, Suzuki Y, Xie Q, Jia J, Karino Y, Hou J, Chayama K, Imamura M, Lao-Tan JY, Lim SG, Tanaka Y, Xie W, Yoon JH, Duan Z, Kurosaki M, Park SJ, Labio ME, Kumar R, Kweon YO, Yim HJ, Tao Y, Cremer J, Elston R, Davies M, Baptiste-Brown S, Han K, Campbell FM, Paff M, Theodore D. Phase IIa, randomised, double-blind study of GSK3389404 in patients with chronic hepatitis B on stable nucleos(t)ide therapy. J Hepatol. 2022 Oct;77(4):967-977. doi: 10.1016/j.jhep.2022.05.031. Epub 2022 Jun 15. PMID 35714812

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2a study examining the first administration of GSK3389404 in participants with chronic hepatitis B (CHB). The study was conducted in 2 parts- Part 1 (dose escalation) and Part 2 (dose expansion and optional follow-up period).
Pre-assignment Details: A total of 106 participants were screened, of which 78 participants (12 participants in Part 1 and 66 participants in Part 2) were enrolled and received either GSK3389404 or placebo. No participants were enrolled in two cohorts of Part 1 (GSK3389404 60 milligram [mg] and GSK3389404 240 mg) as per decision made by the dose escalation committee.
Groups:
- Part 1: Placebo: Participants received a single dose of Placebo via subcutaneous (SC) route on Day 1.
- Part 1: GSK3389404 30 mg: Participants received a single dose of GSK3389404 30 mg via SC route on Day 1.
- Part 1: GSK3389404 60 mg: Participants received a single dose of GSK3389404 60 mg via SC route on Day 1.
- Part 1: GSK3389404 120 mg: Participants received a single dose of GSK3389404 120 mg via SC route on Day 1.
- Part 1: GSK3389404 240 mg: Participants received a single dose of GSK3389404 240 mg via SC route on Day 1.
- Part 2: Placebo: Participants received once weekly SC dose of Placebo until Day 78. Participants who completed Day 169 visit were given an option to enter optional follow-up (FU) period up to Day 450.
- Part 2: GSK3389404 30 mg Weekly: Participants received once weekly SC dose of GSK3389404 30 mg until Day 78. Participants who completed Day 169 visit were given an option to enter optional follow-up (FU) period up to Day 450.
- Part 2: GSK3389404 60 mg Weekly: Participants received once weekly SC dose of GSK3389404 60 mg until Day 78. Participants who completed Day 169 visit were given an option to enter optional follow-up (FU) period up to Day 450.
- Part 2: GSK3389404 120 mg Bi-weekly: Participants received bi-weekly SC dose of GSK3389404 120 mg until Day 71. Participants who completed Day 169 visit were given an option to enter optional follow-up (FU) period up to Day 450.
- Part 2: GSK3389404 120 mg Weekly: Participants received once weekly SC dose of GSK3389404 120 mg until Day 78. Participants who completed Day 169 visit were given an option to enter optional follow-up (FU) period up to Day 450.
Period: Part 1 (Up to 60 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg | Part 1: GSK3389404 240 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Started | 3 | 3 | 0 (No participants were enrolled in this arm as per decision made by the dose escalation committee.) | 6 | 0 (No participants were enrolled in this arm as per decision made by the dose escalation committee.) | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Up to 169 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg | Part 1: GSK3389404 240 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Started | 0 | 0 | 0 | 0 | 0 | 10 | 6 | 20 | 15 | 15
Completed | 0 | 0 | 0 | 0 | 0 | 10 | 6 | 19 | 14 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 2:Optional FU (Up to 450 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg | Part 1: GSK3389404 240 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Started | 0 | 0 | 0 | 0 | 0 | 10 | 5 (1 participant didn't enter into optional follow-up period.) | 17 (2 participants didn't enter into optional follow-up period.) | 13 (1 participant did not enter into optional follow-up period) | 15
Completed | 0 | 0 | 0 | 0 | 0 | 9 | 5 | 17 | 10 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in two cohorts of Part 1 (GSK3389404 60 mg and GSK3389404 240 mg) as per decision made by the dose escalation committee.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly | Total
Number analyzed (Participants) | 3 | 3 | 6 | 10 | 6 | 20 | 15 | 15 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6 | 8 | 5 | 20 | 15 | 15 | 75
  >=65 years | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4 | 1 | 10 | 2 | 2 | 23
  Male | 2 | 3 | 3 | 6 | 5 | 10 | 13 | 13 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian Heritage | 1 | 0 | 3 | 4 | 0 | 9 | 11 | 9 | 37
  Asian-Japanese Heritage | 0 | 0 | 0 | 4 | 6 | 7 | 3 | 5 | 25
  Asian-South East Asian Heritage | 2 | 3 | 3 | 2 | 0 | 4 | 1 | 0 | 15
  Mixed Asian Race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time Points
Description: SBP and DBP were measured in a supine or semi-supine position after approximately 5 minutes rest. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Day 1: 1 hour, Day 1: 2 hours, Day 1: 4 hours, Day 1: 8 hours, Day 3, Day 8 and Day 30
Population: Safety Population comprised of all participants who received at least one dose of the study treatment (including placebo). Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Millimeters of mercury (mmHg)
  DBP, Day 1: 1 hour, n=3,3,6 | -3.67 (16.073) | 3.00 (7.550) | 0.50 (11.554)
  DBP, Day 1: 2 hour, n=3,3,6 | -5.33 (9.018) | -3.33 (3.055) | -4.33 (8.847)
  DBP, Day 1: 4 hour, n=3,3,6 | -8.50 (7.365) | -7.67 (1.528) | -10.50 (6.626)
  DBP, Day 1: 8 hour, n=3,3,6 | -7.17 (16.510) | -0.50 (2.784) | -3.17 (7.414)
  DBP, Day 3, n=3,3,6 | -7.00 (20.075) | -5.83 (5.107) | -2.33 (5.538)
  DBP, Day 8, n=2,3,6: number analyzed (Participants) | 2 | 3 | 6
  DBP, Day 8, n=2,3,6 | -7.50 (20.506) | -1.00 (7.000) | -1.50 (9.731)
  DBP, Day 30, n=3,3,6 | -6.33 (19.604) | -6.00 (1.000) | -3.00 (10.431)
  SBP, Day 1: 1 hour, n=3,3,6 | -0.17 (4.072) | 5.72 (9.595) | -2.33 (16.367)
  SBP, Day 1: 2 hour, n=3,3,6 | -3.83 (17.061) | 6.89 (13.040) | -6.00 (12.083)
  SBP, Day 1: 4 hour, n=3,3,6 | -13.33 (14.012) | 0.06 (6.646) | -8.00 (14.269)
  SBP, Day 1: 8 hour, n=3,3,6 | -5.50 (13.611) | 0.89 (4.550) | -5.67 (12.644)
  SBP, Day 3, n=3,3,6 | -3.00 (21.633) | -7.94 (3.084) | -0.83 (9.261)
  SBP, Day 8, n=2,3,6: number analyzed (Participants) | 2 | 3 | 6
  SBP, Day 8, n=2,3,6 | 6.00 (32.527) | 4.06 (5.149) | 0.17 (4.070)
  SBP, Day 30, n=3,3,6 | -2.00 (26.514) | 4.89 (12.303) | 3.67 (13.736)

2. Primary Outcome: Part 2: Change From Baseline in SBP and DBP at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 1
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
mmHg
  DBP, Day 8, n=10,6,20,15,15 | 5.8 (8.90) | 2.3 (8.71) | -1.9 (7.13) | 1.0 (8.86) | -0.7 (8.61)
  DBP, Day 15, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 15, n=10,6,20,14,15 | 2.1 (8.46) | -4.0 (13.02) | -0.3 (9.09) | -0.3 (7.09) | -2.7 (7.32)
  DBP, Day 22, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 22, n=10,6,20,14,15 | 3.4 (9.49) | -2.0 (6.20) | 0.3 (8.77) | 1.6 (9.80) | -3.0 (9.13)
  DBP, Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  DBP, Day 29, n=10,6,20,13,15 | 3.9 (8.77) | 3.3 (2.25) | -1.7 (8.55) | 2.1 (9.71) | -0.7 (7.35)
  DBP, Day 36, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 36, n=10,6,20,14,15 | 1.8 (8.90) | -1.7 (9.35) | -0.8 (8.84) | 1.9 (8.46) | -0.1 (6.38)
  DBP, Day 43, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 43, n=10,6,20,14,15 | 4.2 (12.33) | 0.0 (6.45) | -0.3 (12.38) | 0.9 (10.99) | -0.8 (6.12)
  DBP, Day 50, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  DBP, Day 50, n=10,6,19,14,15 | 11.0 (17.26) | 2.8 (8.93) | 0.1 (9.95) | 1.3 (10.25) | -3.2 (7.74)
  DBP, Day 57, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 57, n=10,6,20,14,15 | 4.0 (9.88) | -0.2 (8.73) | -0.5 (9.10) | 1.6 (8.34) | -0.8 (8.16)
  DBP, Day 64, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 64, n=10,6,20,14,15 | 3.2 (9.67) | 0.3 (9.31) | -1.9 (10.27) | 2.1 (9.71) | -1.8 (9.93)
  DBP, Day 71, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 71, n=10,6,20,14,15 | 2.9 (9.56) | 3.8 (7.11) | -0.6 (9.83) | 3.1 (9.92) | 1.4 (9.74)
  DBP, Day 78, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 78, n=10,6,20,14,15 | 4.6 (5.50) | 1.2 (6.59) | -0.8 (8.80) | 5.0 (8.71) | -4.2 (9.85)
  DBP, Day 85, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 85, n=10,6,20,14,15 | 4.9 (7.20) | 1.0 (9.47) | -1.2 (12.35) | 6.4 (11.21) | -2.3 (10.69)
  DBP, Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  DBP, Day 92, n=10,6,19,14,15 | 2.9 (7.39) | 3.8 (7.63) | -2.2 (9.52) | 3.9 (9.08) | -1.1 (10.00)
  DBP, Day 99, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 99, n=10,6,20,14,15 | 4.3 (10.27) | 3.0 (9.86) | 0.3 (10.80) | 1.3 (10.38) | 0.1 (10.80)
  DBP, Day 113, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 113, n=10,6,20,14,15 | 5.9 (9.71) | 2.7 (8.80) | -1.2 (10.96) | 4.9 (8.28) | 2.9 (8.17)
  DBP, Day 141, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  DBP, Day 141, n=10,6,20,14,15 | 7.5 (10.20) | 1.2 (8.33) | 0.7 (12.37) | 0.8 (8.51) | 1.1 (11.28)
  DBP, Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  DBP, Day 169, n=10,6,19,14,15 | 5.8 (10.13) | 6.3 (11.71) | 0.5 (11.14) | 3.4 (12.07) | -0.3 (8.83)
  SBP, Day 8, n=10,6,20,15,15 | 7.7 (11.17) | 5.0 (7.40) | -2.6 (10.45) | 0.8 (14.35) | 2.1 (9.59)
  SBP, Day 15, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 15, n=10,6,20,14,15 | 8.0 (11.60) | 1.7 (14.42) | -0.4 (10.02) | 2.1 (12.77) | 0.1 (11.03)
  SBP, Day 22, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 22, n=10,6,20,14,15 | 5.7 (13.72) | 1.5 (6.57) | -2.2 (8.66) | 2.4 (11.54) | -2.1 (14.36)
  SBP, Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  SBP, Day 29, n=10,6,20,13,15 | 6.1 (13.20) | 1.7 (4.27) | -3.1 (11.83) | 2.9 (16.89) | 1.5 (10.29)
  SBP, Day 36, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 36, n=10,6,20,14,15 | 0.2 (11.43) | -0.5 (12.05) | -5.6 (10.54) | 0.4 (16.21) | 2.1 (12.90)
  SBP, Day 43, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 43, n=10,6,20,14,15 | 5.6 (9.91) | 4.7 (13.22) | -0.6 (11.89) | 1.7 (16.11) | 0.0 (12.53)
  SBP, Day 50, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  SBP, Day 50, n=10,6,19,14,15 | 5.2 (14.88) | 4.7 (9.65) | -3.4 (11.93) | 1.6 (12.74) | -2.2 (11.36)
  SBP, Day 57, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 57, n=10,6,20,14,15 | 1.7 (13.86) | 2.5 (13.40) | -4.2 (10.21) | 0.1 (14.91) | 0.9 (17.26)
  SBP, Day 64, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 64, n=10,6,20,14,15 | 5.1 (11.98) | 0.2 (9.11) | -4.1 (9.17) | 1.4 (16.29) | 0.5 (15.50)
  SBP, Day 71, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 71, n=10,6,20,14,15 | 4.6 (11.98) | 5.0 (10.22) | -2.2 (11.97) | 4.8 (17.68) | 4.2 (12.46)
  SBP, Day 78, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 78, n=10,6,20,14,15 | 5.2 (12.28) | 5.0 (6.16) | -4.4 (10.09) | 4.1 (13.95) | -0.1 (12.99)
  SBP, Day 85, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 85, n=10,6,20,14,15 | 7.2 (15.22) | 5.2 (9.06) | -5.0 (12.73) | 6.2 (15.62) | -3.5 (14.30)
  SBP, Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  SBP, Day 92, n=10,6,19,14,15 | 5.0 (12.57) | 4.3 (8.50) | -4.1 (12.60) | 4.6 (13.87) | -0.1 (12.14)
  SBP, Day 99, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 99, n=10,6,20,14,15 | 7.1 (16.84) | 3.3 (15.45) | -0.5 (14.05) | 1.6 (16.46) | 2.2 (16.34)
  SBP, Day 113, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 113, n=10,6,20,14,15 | 7.3 (13.30) | 5.7 (9.35) | -3.2 (11.64) | 4.9 (12.07) | 6.6 (10.72)
  SBP, Day 141, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  SBP, Day 141, n=10,6,20,14,15 | 10.9 (11.51) | 3.5 (9.81) | -0.9 (12.77) | 2.9 (15.93) | 4.6 (16.85)
  SBP, Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  SBP, Day 169, n=10,6,19,14,15 | 11.8 (12.41) | 9.7 (12.45) | 0.8 (11.61) | 5.1 (17.41) | 4.9 (12.85)

3. Primary Outcome: Part 2: Change From Baseline in SBP and DBP at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: as for outcome 1
Time Frame: Baseline (Day 1 pre-dose), Day 270 and Day 450
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
mmHg
  DBP, Day 270, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  DBP, Day 270, n=1,0,0,0,0 | -9.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |  |  |
  DBP, Day 450, n=0,0,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  DBP, Day 450, n=0,0,1,0,0 |  |  | 7.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |
  SBP, Day 270, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  SBP, Day 270, n=1,0,0,0,0 | -18.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |  |  |
  SBP, Day 450, n=0,0,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  SBP, Day 450, n=0,0,1,0,0 |  |  | 3.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |

4. Primary Outcome: Part 1: Change From Baseline in Heart Rate at Indicated Time Points
Description: Heart rate was measured in a supine or semi-supine position after approximately 5 minutes rest. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Day 1: 1 hour, Day 1: 2 hours, Day 1: 4 hours, Day 1: 8 hours, Day 3, Day 8 and Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Beats per minute
  Day 1: 1 hour, n=3,3,6 | 4.78 (3.977) | 1.44 (8.694) | -5.00 (2.530)
  Day 1: 2 hour, n=3,3,6 | 13.94 (12.537) | 4.61 (17.472) | -2.17 (6.338)
  Day 1: 4 hour, n=3,3,6 | 8.11 (3.564) | -0.22 (16.201) | -0.17 (7.055)
  Day 1: 8 hour, n=3,3,6 | 5.61 (5.029) | -5.22 (15.827) | -0.17 (3.430)
  Day 3, n=3,3,6 | 12.11 (4.439) | 2.11 (3.657) | 2.50 (9.503)
  Day 8, n=2,3,6: number analyzed (Participants) | 2 | 3 | 6
  Day 8, n=2,3,6 | 8.00 (4.243) | -2.89 (13.104) | 2.00 (10.863)
  Day 30, n=3,3,6 | 6.44 (16.194) | 3.28 (14.958) | 1.50 (10.134)

5. Primary Outcome: Part 2: Change From Baseline in Heart Rate at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 4
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Beats per minute
  Day 8, n=10,6,20,15,15 | 9.9 (9.22) | 6.2 (9.15) | 2.8 (9.92) | 5.7 (8.96) | 5.2 (8.97)
  Day 15, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 15, n=10,6,20,14,15 | 9.2 (13.89) | -3.0 (6.90) | 3.6 (10.64) | 2.1 (6.92) | 2.3 (9.54)
  Day 22, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 22, n=10,6,20,14,15 | 6.3 (13.53) | 4.7 (7.89) | 3.8 (11.57) | 2.6 (7.78) | 1.6 (9.52)
  Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, n=10,6,20,13,15 | 5.5 (11.32) | 3.5 (7.92) | 1.2 (10.25) | 1.8 (8.99) | 1.3 (6.84)
  Day 36, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 36, n=10,6,20,14,15 | 7.8 (10.99) | 5.7 (11.69) | 2.1 (7.32) | 4.0 (9.97) | 1.5 (8.70)
  Day 43, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 43, n=10,6,20,14,15 | 5.1 (13.76) | 5.0 (11.03) | 2.8 (12.53) | 3.0 (11.57) | 4.8 (9.92)
  Day 50, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 50, n=10,6,19,14,15 | 7.9 (12.52) | 5.3 (11.38) | 2.6 (10.89) | 4.6 (11.47) | 1.5 (9.85)
  Day 57, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 57, n=10,6,20,14,15 | 2.9 (12.78) | -4.0 (11.01) | 1.1 (10.19) | 2.1 (8.39) | 1.1 (8.33)
  Day 64, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 64, n=10,6,20,14,15 | 5.1 (13.24) | -1.2 (9.43) | 3.0 (10.50) | 4.5 (11.35) | 1.9 (7.90)
  Day 71, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 71, n=10,6,20,14,15 | 4.8 (14.30) | -2.2 (9.58) | 4.7 (12.01) | 0.6 (9.70) | 2.5 (9.13)
  Day 78, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 78, n=10,6,20,14,15 | 3.9 (13.70) | 0.2 (10.80) | 5.5 (10.31) | 2.4 (6.59) | 3.0 (7.63)
  Day 85, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 85, n=10,6,20,14,15 | 7.2 (15.30) | -0.2 (10.38) | 3.6 (10.63) | 1.4 (8.04) | 0.5 (9.56)
  Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 92, n=10,6,19,14,15 | 6.4 (14.01) | 1.2 (8.95) | 4.6 (10.23) | 4.3 (10.29) | 0.5 (9.23)
  Day 99, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 99, n=10,6,20,14,15 | 3.9 (11.93) | 6.7 (11.27) | 4.0 (12.09) | 2.5 (8.23) | 4.5 (10.59)
  Day 113, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 113, n=10,6,20,14,15 | 7.5 (15.92) | 3.8 (9.33) | 1.5 (9.14) | 3.6 (6.50) | 4.8 (8.54)
  Day 141, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 141, n=10,6,20,14,15 | 5.7 (16.89) | 0.8 (14.74) | 3.4 (8.32) | 5.1 (8.77) | 4.3 (10.22)
  Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, n=10,6,19,14,15 | 7.9 (16.31) | 2.8 (13.04) | 4.3 (9.59) | 4.7 (8.72) | 3.1 (6.75)

6. Primary Outcome: Part 2: Change From Baseline in Heart Rate at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: as for outcome 4
Time Frame: Baseline (Day 1 pre-dose), Day 270 and Day 450
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
Beats per minute
  Day 270, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 270, n=1,0,0,0,0 | -26.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |  |  |
  Day 450, n=0,0,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Day 450, n=0,0,1,0,0 |  |  | -11.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |

7. Primary Outcome: Part 1: Change From Baseline in Respiratory Rate at Indicated Time Points
Description: Respiratory rate was measured in a supine or semi-supine position after approximately 5 minutes rest. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Days 3, 8 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Breaths per minute
  Day 3, n=3,3,6 | -0.67 (0.577) | -1.00 (1.732) | -0.33 (1.862)
  Day 8, n=2,3,6: number analyzed (Participants) | 2 | 3 | 6
  Day 8, n=2,3,6 | -0.50 (0.707) | -1.00 (1.000) | 0.00 (2.280)
  Day 30, n=3,3,6 | -1.33 (1.155) | -0.67 (1.528) | 0.50 (2.258)

8. Primary Outcome: Part 2: Change From Baseline in Respiratory Rate at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 7
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Breaths per minute
  Day 8, n=10,6,20,15,15 | 0.00 (1.94) | -0.8 (4.49) | 0.5 (1.82) | -0.3 (1.35) | -0.3 (1.94)
  Day 15, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 15, n=10,6,20,14,15 | -0.2 (2.25) | -1.3 (5.28) | -0.1 (0.91) | -0.3 (1.64) | -0.6 (2.53)
  Day 22, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 22, n=10,6,20,14,15 | 0.1 (2.77) | -1.3 (5.28) | 0.6 (1.36) | -0.4 (1.28) | -0.2 (1.74)
  Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, n=10,6,20,13,15 | -0.6 (2.37) | 0.2 (3.71) | -0.7 (2.49) | -0.9 (1.61) | -0.7 (2.23)
  Day 36, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 36, n=10,6,20,14,15 | -0.3 (3.27) | -0.8 (5.00) | 0.6 (1.23) | -0.7 (1.49) | 0.2 (1.90)
  Day 43, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 43, n=10,6,20,14,15 | 0.0 (2.36) | -0.8 (5.00) | 0.2 (1.46) | -0.3 (1.27) | -0.1 (1.41)
  Day 50, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 50, n=10,6,19,14,15 | -0.2 (2.44) | -1.0 (5.51) | 0.4 (1.07) | -0.5 (1.34) | 0.1 (1.39)
  Day 57, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 57, n=10,6,20,14,15 | -0.3 (3.09) | 0.0 (3.85) | 0.5 (1.64) | 0.0 (1.04) | 0.2 (2.54)
  Day 64, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 64, n=10,6,20,14,15 | 0.0 (2.45) | -0.7 (4.89) | 0.4 (1.10) | -0.3 (1.27) | 0.2 (1.74)
  Day 71, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 71, n=10,6,20,14,15 | -0.1 (2.38) | -0.7 (4.89) | 0.2 (1.24) | -0.2 (1.31) | 0.4 (1.50)
  Day 78, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 78, n=10,6,20,14,15 | 0.2 (2.78) | -1.0 (5.51) | 0.5 (1.50) | 0.3 (1.64) | -0.7 (2.06)
  Day 85, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 85, n=10,6,20,14,15 | 0.4 (2.63) | -0.8 (5.19) | 0.3 (1.63) | 0.1 (1.49) | 0.0 (1.31)
  Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 92, n=10,6,19,14,15 | 0.4 (2.01) | -1.3 (5.50) | 0.1 (1.37) | -0.4 (1.79) | 0.3 (1.29)
  Day 99, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 99, n=10,6,20,14,15 | 0.2 (2.15) | -1.0 (4.29) | -0.1 (1.85) | 0.1 (1.54) | 0.5 (1.46)
  Day 113, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 113, n=10,6,20,14,15 | 0.7 (3.09) | -1.0 (4.90) | 0.3 (1.38) | -0.1 (1.44) | 0.0 (1.93)
  Day 141, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 141, n=10,6,20,14,15 | 0.5 (3.27) | -1.0 (4.90) | 0.4 (1.19) | -0.2 (1.42) | -0.1 (2.03)
  Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, n=10,6,19,14,15 | 0.1 (2.69) | -1.0 (4.90) | 0.6 (1.30) | 0.0 (1.36) | 0.1 (2.15)

9. Primary Outcome: Part 2: Change From Baseline in Respiratory Rate at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: as for outcome 7
Time Frame: Baseline (Day 1 pre-dose), Day 270 and Day 450
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
Breaths per minute
  Day 270, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 270, n=1,0,0,0,0 | 0.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |  |  |
  Day 450, n=0,0,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Day 450, n=0,0,1,0,0 |  |  | 2.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |

10. Primary Outcome: Part 1: Change From Baseline in Body Temperature at Indicated Time Points
Description: Body temperature was measured in a supine or semi-supine position after approximately 5 minutes rest. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Days 3, 8 and 30
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Degrees Celsius
  Day 3, n=3,3,6 | 0.10 (0.100) | 0.37 (0.306) | 0.25 (0.345)
  Day 8, n=2,3,6: number analyzed (Participants) | 2 | 3 | 6
  Day 8, n=2,3,6 | 0.20 (0.283) | -0.03 (0.351) | 0.08 (0.343)
  Day 30, n=3,3,6 | 0.10 (0.173) | 0.20 (0.361) | 0.10 (0.358)

11. Primary Outcome: Part 2: Change From Baseline in Body Temperature at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 10
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Degrees Celsius
  Day 8, n=10,6,20,15,15 | 0.24 (0.366) | -0.02 (0.366) | 0.18 (0.466) | -0.15 (0.385) | -0.11 (0.337)
  Day 15, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 15, n=10,6,20,14,15 | 0.18 (0.447) | -0.12 (0.397) | 0.07 (0.443) | -0.07 (0.350) | 0.08 (0.428)
  Day 22, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 22, n=10,6,20,14,15 | 0.01 (0.692) | 0.07 (0.344) | 0.06 (0.491) | 0.05 (0.277) | -0.09 (0.350)
  Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, n=10,6,20,13,15 | 0.21 (0.370) | -0.13 (0.423) | 0.19 (0.433) | 0.00 (0.430) | 0.05 (0.505)
  Day 36, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 36, n=10,6,20,14,15 | 0.25 (0.354) | 0.15 (0.266) | 0.15 (0.501) | -0.09 (0.421) | -0.10 (0.606)
  Day 43, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 43, n=10,6,20,14,15 | 0.10 (0.365) | 0.05 (0.243) | 0.25 (0.399) | -0.15 (0.313) | -0.04 (0.557)
  Day 50, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 50, n=10,6,19,14,15 | 0.12 (0.609) | 0.07 (0.258) | 0.26 (0.352) | -0.12 (0.428) | -0.07 (0.746)
  Day 57, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 57, n=10,6,20,14,15 | 0.06 (0.395) | 0.02 (0.366) | 0.15 (0.380) | -0.06 (0.332) | 0.07 (0.575)
  Day 64, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 64, n=10,6,20,14,15 | 0.07 (0.581) | -0.03 (0.301) | 0.17 (0.386) | -0.04 (0.393) | -0.01 (0.536)
  Day 71, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 71, n=10,6,20,14,15 | 0.26 (0.599) | -0.25 (0.207) | 0.26 (0.425) | -0.14 (0.413) | 0.08 (0.684)
  Day 78, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 78, n=10,6,20,14,15 | 0.14 (0.450) | -0.13 (0.216) | 0.20 (0.349) | -0.08 (0.283) | 0.00 (0.679)
  Day 85, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 85, n=10,6,20,14,15 | 0.19 (0.716) | 0.08 (0.240) | 0.25 (0.412) | -0.09 (0.398) | 0.04 (0.622)
  Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 92, n=10,6,19,14,15 | -0.11 (0.729) | -0.07 (0.280) | 0.24 (0.356) | -0.14 (0.337) | 0.01 (0.645)
  Day 99, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 99, n=10,6,20,14,15 | 0.16 (0.443) | 0.15 (0.259) | 0.26 (0.378) | -0.13 (0.305) | -0.04 (0.505)
  Day 113, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 113, n=10,6,20,14,15 | 0.03 (0.397) | 0.05 (0.281) | 0.20 (0.419) | -0.03 (0.327) | -0.10 (0.535)
  Day 141, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 141, n=10,6,20,14,15 | 0.14 (0.556) | -0.13 (0.320) | 0.14 (0.547) | -0.19 (0.366) | -0.03 (0.635)
  Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, n=10,6,19,14,15 | 0.12 (0.592) | -0.08 (0.240) | 0.21 (0.494) | -0.02 (0.412) | 0.04 (0.612)

12. Primary Outcome: Part 2: Change From Baseline in Body Temperature at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: as for outcome 10
Time Frame: Baseline (Day 1 pre-dose), Day 270 and Day 450
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
Degrees Celsius
  Day 270, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Day 270, n=1,0,0,0,0 | -0.40 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |  |  |
  Day 450, n=0,0,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Day 450, n=0,0,1,0,0 |  |  | 0.40 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant. |  |

13. Primary Outcome: Part 1: Number of Participants With Abnormal Findings in Physical Examination
Description: Physical examinations included assessment of the dermatologic, cardiovascular, respiratory, gastrointestinal, and neurological systems. Data was not collected and not captured in the database.
Time Frame: Up to Day 60
Population: Safety Population. Data was not collected and not captured in the database.
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0

14. Primary Outcome: Part 2: Number of Participants With Abnormal Findings in Physical Examination (Up to Day 169-Interim Analysis)
Description: as for outcome 13
Time Frame: Up to Day 169
Population: Safety Population. Data was not collected and not captured in the database.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Part 2: Number of Participants With Abnormal Findings in Physical Examination (Up to Day 450-Optional Follow-up)
Description: as for outcome 13
Time Frame: Up to Day 450
Population: Safety Population. Data was not collected and not captured in the database.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Part 1: Number of Participants With Maximum Post-Baseline Grade by Category in Hematology and Coagulation Parameters
Description: Blood samples were collected for the analysis of following hematology and coagulation parameters: Hemoglobin, Leukocytes, Lymphocytes, Neutrophils, Platelets, Activated partial thromboplastin time (aPTT), Prothrombin international normalized ratio (INR) and Prothrombin time (PT). Laboratory parameters were graded according to Division of Acquired Immune Deficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Only those hematology and coagulation parameters with maximum post-Baseline grade (Grade 1 to Grade 4) have been presented.
Time Frame: Up to Day 60
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants
  Hemoglobin, Grade 1 | 0 | 0 | 0
  Hemoglobin, Grade 2 | 0 | 0 | 0
  Hemoglobin, Grade 3 | 0 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0 | 0
  Leukocyte, Grade 1 | 0 | 0 | 0
  Leukocyte, Grade 2 | 0 | 0 | 0
  Leukocyte, Grade 3 | 0 | 0 | 0
  Leukocyte, Grade 4 | 0 | 0 | 0
  Lymphocyte, Grade 1 | 0 | 0 | 0
  Lymphocyte, Grade 2 | 0 | 0 | 1
  Lymphocyte, Grade 3 | 0 | 0 | 0
  Lymphocyte, Grade 4 | 0 | 0 | 0
  Neutrophil, Grade 1 | 0 | 0 | 0
  Neutrophil, Grade 2 | 0 | 0 | 0
  Neutrophil, Grade 3 | 0 | 0 | 0
  Neutrophil, Grade 4 | 0 | 0 | 0
  Platelet, Grade 1 | 0 | 0 | 0
  Platelet, Grade 2 | 0 | 0 | 0
  Platelet, Grade 3 | 0 | 0 | 0
  Platelet, Grade 4 | 0 | 0 | 0
  aPTT, Grade 1 | 1 | 1 | 1
  aPTT, Grade 2 | 0 | 0 | 0
  aPTT, Grade 3 | 0 | 0 | 0
  aPTT, Grade 4 | 0 | 0 | 0
  Prothrombin INR, Grade 1 | 0 | 0 | 0
  Prothrombin INR, Grade 2 | 0 | 0 | 0
  Prothrombin INR, Grade 3 | 0 | 0 | 0
  Prothrombin INR, Grade 4 | 0 | 0 | 0
  PT, Grade 1 | 0 | 0 | 1
  PT, Grade 2 | 0 | 0 | 0
  PT, Grade 3 | 0 | 0 | 0
  PT, Grade 4 | 0 | 0 | 0

17. Primary Outcome: Part 2: Number of Participants With Maximum Post-Baseline Grade by Category in Hematology and Coagulation Parameters (Up to Day 169-Interim Analysis)
Description: Blood samples were collected for the analysis of following hematology and coagulation parameters: Hemoglobin, Leukocytes, Lymphocytes, Neutrophils, Platelets, aPTT, Prothrombin INR and PT. Laboratory parameters were graded according to DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Only those hematology and coagulation parameters with maximum post-Baseline grade (Grade 1 to Grade 4) have been presented.
Time Frame: Up to Day 169
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Participants
  Hemoglobin, Grade 1 | 0 | 1 | 0 | 0 | 0
  Hemoglobin, Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0 | 0 | 0 | 0
  Leukocyte, Grade 1 | 0 | 0 | 0 | 1 | 1
  Leukocyte, Grade 2 | 0 | 0 | 0 | 0 | 0
  Leukocyte, Grade 3 | 0 | 0 | 0 | 0 | 0
  Leukocyte, Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte, Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte, Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte, Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte, Grade 4 | 0 | 0 | 0 | 0 | 0
  Neutrophil, Grade 1 | 0 | 0 | 0 | 1 | 3
  Neutrophil, Grade 2 | 0 | 0 | 0 | 0 | 0
  Neutrophil, Grade 3 | 0 | 0 | 0 | 0 | 0
  Neutrophil, Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelet, Grade 1 | 0 | 0 | 1 | 0 | 2
  Platelet, Grade 2 | 0 | 0 | 0 | 0 | 1
  Platelet, Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet, Grade 4 | 0 | 0 | 0 | 0 | 0
  aPTT, Grade 1 | 1 | 2 | 5 | 4 | 5
  aPTT, Grade 2 | 0 | 0 | 0 | 0 | 1
  aPTT, Grade 3 | 0 | 0 | 0 | 0 | 0
  aPTT, Grade 4 | 0 | 0 | 0 | 0 | 0
  Prothrombin INR, Grade 1 | 0 | 0 | 3 | 0 | 1
  Prothrombin INR, Grade 2 | 0 | 0 | 0 | 0 | 1
  Prothrombin INR, Grade 3 | 0 | 0 | 0 | 0 | 0
  Prothrombin INR, Grade 4 | 0 | 0 | 0 | 0 | 0
  PT, Grade 1 | 0 | 0 | 6 | 0 | 5
  PT, Grade 2 | 0 | 0 | 0 | 0 | 0
  PT, Grade 3 | 0 | 0 | 0 | 0 | 1
  PT, Grade 4 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Part 2: Number of Participants With Maximum Post-Baseline Grade by Category in Hematology and Coagulation Parameters (Up to Day 450-Optional Follow-up)
Description: as for outcome 17
Time Frame: Up to Day 450
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Participants
  Hemoglobin, Grade 1 | 0 | 1 | 0 | 0 | 0
  Hemoglobin, Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0 | 0 | 0 | 0
  Leukocyte, Grade 1 | 0 | 0 | 0 | 1 | 1
  Leukocyte, Grade 2 | 0 | 0 | 0 | 0 | 0
  Leukocyte, Grade 3 | 0 | 0 | 0 | 0 | 0
  Leukocyte, Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte, Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte, Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte, Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte, Grade 4 | 0 | 0 | 0 | 0 | 0
  Neutrophil, Grade 1 | 0 | 0 | 0 | 1 | 3
  Neutrophil, Grade 2 | 0 | 0 | 0 | 0 | 0
  Neutrophil, Grade 3 | 0 | 0 | 0 | 0 | 0
  Neutrophil, Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelet, Grade 1 | 0 | 0 | 1 | 0 | 2
  Platelet, Grade 2 | 0 | 0 | 0 | 0 | 1
  Platelet, Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet, Grade 4 | 0 | 0 | 0 | 0 | 0
  aPTT, Grade 1 | 1 | 2 | 5 | 4 | 5
  aPTT, Grade 2 | 0 | 0 | 0 | 0 | 1
  aPTT, Grade 3 | 0 | 0 | 0 | 0 | 0
  aPTT, Grade 4 | 0 | 0 | 0 | 0 | 0
  Prothrombin INR, Grade 1 | 0 | 0 | 3 | 0 | 1
  Prothrombin INR, Grade 2 | 0 | 0 | 0 | 0 | 1
  Prothrombin INR, Grade 3 | 0 | 0 | 0 | 0 | 0
  Prothrombin INR, Grade 4 | 0 | 0 | 0 | 0 | 0
  PT, Grade 1 | 0 | 1 | 6 | 0 | 5
  PT, Grade 2 | 0 | 0 | 0 | 0 | 0
  PT, Grade 3 | 0 | 0 | 0 | 0 | 1
  PT, Grade 4 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Part 1: Change From Baseline in Complement C3 and Complement C4 Level at Indicated Time Points
Description: Blood samples were collected from participants to assess complement C3 and complement C4 levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Milligram per deciliter
  Complement C3 | -8.7 (11.24) | -13.0 (3.00) | -16.3 (7.74)
  Complement C4 | -2.0 (2.00) | -2.3 (0.58) | -4.2 (3.76)

20. Primary Outcome: Part 2: Change From Baseline in Complement C3 and Complement C4 Level at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 19
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 169
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Milligram per deciliter
  Complement C3 | -11.0 (16.10) | -13.5 (9.14) | -11.3 (10.38) | -10.9 (15.19) | -17.7 (13.98)
  Complement C4 | -3.5 (2.12) | -4.7 (4.41) | -3.8 (2.57) | -3.4 (2.13) | -5.6 (3.07)

21. Primary Outcome: Part 2: Change From Baseline in Complement C3 and Complement C4 Level at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Blood samples were planned to be collected from participants to evaluate change from Baseline in complement C3 and complement C4 levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was to be calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: Safety Population. Data was not collected for this outcome measure during optional follow-up period.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: Part 1: Change From Baseline in Complement Bb Level at Indicated Time Points
Description: Blood samples were collected from participants to assess complement Bb levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligram per liter
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Milligram per liter | 0.193 (0.2409) | 0.023 (0.0950) | 0.150 (0.2119)

23. Primary Outcome: Part 2: Change From Baseline in Complement Bb Level at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 22
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 169
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligram per liter
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Milligram per liter | 0.245 (0.319) | 0.198 (0.143) | 0.315 (0.740) | 0.115 (0.222) | -0.007 (0.30)

24. Primary Outcome: Part 2: Change From Baseline in Complement Bb Level at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Blood samples were collected from participants to evaluate change from Baseline in complement Bb levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligram per liter
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Milligram per liter | 0.304 (0.295) | 0.365 (0.269) | 0.436 (0.679) | 0.173 (0.213) | 0.107 (0.367)

25. Primary Outcome: Part 1: Change From Baseline in Complement C5a Level at Indicated Time Points
Description: Blood samples were collected from participants to assess complement C5a levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Microgram per liter
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Microgram per liter | 1.497 (0.6306) | 0.373 (0.9952) | -1.267 (5.7581)

26. Primary Outcome: Part 2: Change From Baseline in Complement C5a Level at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 25
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 169
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Microgram per liter
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Microgram per liter | 1.112 (1.481) | 0.860 (1.625) | 1.781 (2.524) | 0.353 (1.323) | -0.093 (1.54)

27. Primary Outcome: Part 2: Change From Baseline in Complement C5a Level at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Blood samples were collected from participants to evaluate change from Baseline in complement C5a levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Milligrams per liter | 1.324 (1.415) | 2.053 (3.456) | 2.040 (2.481) | 0.470 (1.205) | 0.567 (1.354)

28. Primary Outcome: Part 1: Number of Participants With Maximum Post-Baseline Grade by Category in Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: Alanine aminotransferase, Albumin, Alkaline phosphatase, Aspartate aminotransferase, Bilirubin, Calcium (high), Calcium (low), Creatine kinase, Creatinine, Glucose (high), Glucose (low), Magnesium, Phosphate, Potassium (high), Potassium (low), Sodium (high), Sodium (low) and Urate. Laboratory parameters were graded according to DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Only those clinical chemistry parameters with maximum post-Baseline grade (Grade 1 to Grade 4) have been presented.
Time Frame: Up to Day 60
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants
  Alanine aminotransferase, Grade 1 | 0 | 0 | 0
  Alanine aminotransferase, Grade 2 | 0 | 0 | 1
  Alanine aminotransferase, Grade 3 | 0 | 0 | 0
  Alanine aminotransferase, Grade 4 | 0 | 0 | 0
  Albumin, Grade 1 | 0 | 0 | 0
  Albumin, Grade 2 | 0 | 0 | 0
  Albumin, Grade 3 | 0 | 0 | 0
  Albumin, Grade 4 | 0 | 0 | 0
  Alkaline phosphatase, Grade 1 | 0 | 0 | 0
  Alkaline phosphatase, Grade 2 | 0 | 0 | 0
  Alkaline phosphatase, Grade 3 | 0 | 0 | 0
  Alkaline phosphatase, Grade 4 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 1 | 0 | 0 | 1
  Aspartate aminotransferase, Grade 2 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 3 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 4 | 0 | 0 | 0
  Bilirubin, Grade 1 | 0 | 1 | 1
  Bilirubin, Grade 2 | 0 | 0 | 0
  Bilirubin, Grade 3 | 0 | 0 | 0
  Bilirubin, Grade 4 | 0 | 0 | 0
  Calcium (high), Grade 1 | 0 | 0 | 1
  Calcium (high), Grade 2 | 0 | 0 | 0
  Calcium (high), Grade 3 | 0 | 0 | 0
  Calcium (high), Grade 4 | 0 | 0 | 0
  Calcium (low), Grade 1 | 0 | 0 | 0
  Calcium (low), Grade 2 | 0 | 0 | 0
  Calcium (low), Grade 3 | 0 | 0 | 0
  Calcium (low), Grade 4 | 0 | 0 | 0
  Creatine kinase, Grade 1 | 0 | 1 | 0
  Creatine kinase, Grade 2 | 0 | 0 | 0
  Creatine kinase, Grade 3 | 0 | 0 | 0
  Creatine kinase, Grade 4 | 0 | 0 | 0
  Creatinine, Grade 1 | 0 | 0 | 0
  Creatinine, Grade 2 | 0 | 0 | 0
  Creatinine, Grade 3 | 0 | 0 | 0
  Creatinine, Grade 4 | 0 | 0 | 0
  Glucose (high), Grade 1 | 0 | 0 | 1
  Glucose (high), Grade 2 | 0 | 0 | 0
  Glucose (high), Grade 3 | 0 | 0 | 0
  Glucose (high), Grade 4 | 0 | 0 | 0
  Glucose (low), Grade 1 | 0 | 0 | 0
  Glucose (low), Grade 2 | 0 | 0 | 0
  Glucose (low), Grade 3 | 0 | 0 | 0
  Glucose (low), Grade 4 | 0 | 0 | 0
  Magnesium, Grade 1 | 0 | 0 | 0
  Magnesium, Grade 2 | 0 | 0 | 0
  Magnesium, Grade 3 | 0 | 0 | 0
  Magnesium, Grade 4 | 0 | 0 | 0
  Phosphate, Grade 1 | 0 | 0 | 0
  Phosphate, Grade 2 | 0 | 0 | 0
  Phosphate, Grade 3 | 0 | 0 | 0
  Phosphate, Grade 4 | 0 | 0 | 0
  Potassium (high), Grade 1 | 0 | 0 | 0
  Potassium (high), Grade 2 | 0 | 0 | 0
  Potassium (high), Grade 3 | 0 | 0 | 0
  Potassium (high), Grade 4 | 0 | 0 | 0
  Potassium (low), Grade 1 | 0 | 0 | 0
  Potassium (low), Grade 2 | 0 | 0 | 0
  Potassium (low), Grade 3 | 0 | 0 | 0
  Potassium (low), Grade 4 | 0 | 0 | 0
  Sodium (high), Grade 1 | 0 | 0 | 0
  Sodium (high), Grade 2 | 0 | 0 | 0
  Sodium (high), Grade 3 | 0 | 0 | 0
  Sodium (high), Grade 4 | 0 | 0 | 0
  Sodium (low), Grade 1 | 0 | 0 | 0
  Sodium (low), Grade 2 | 0 | 0 | 0
  Sodium (low), Grade 3 | 0 | 0 | 0
  Sodium (low), Grade 4 | 0 | 0 | 0
  Urate, Grade 1 | 0 | 1 | 0
  Urate, Grade 2 | 0 | 0 | 0
  Urate, Grade 3 | 0 | 0 | 0
  Urate, Grade 4 | 0 | 0 | 0

29. Primary Outcome: Part 2: Number of Participants With Maximum Post-Baseline Grade by Category in Clinical Chemistry Parameters (Up to Day 169-Interim Analysis)
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: Alanine aminotransferase, Albumin, Alkaline phosphatase, Aspartate aminotransferase, Bilirubin, Calcium (high), Calcium (low), Creatine kinase, Creatinine, Glucose (high), Glucose (low), Magnesium, Phosphate, Potassium (high), Potassium (low), Sodium (high), Sodium (low), Urate and glomerular filtration rate (GFR). Laboratory parameters were graded according to DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Only those clinical chemistry parameters with maximum post-Baseline grade (Grade 1 to Grade 4) have been presented.
Time Frame: Up to Day 169
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Participants
  Alanine aminotransferase, Grade 1 | 1 | 0 | 2 | 0 | 4
  Alanine aminotransferase, Grade 2 | 0 | 0 | 0 | 1 | 1
  Alanine aminotransferase, Grade 3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase, Grade 4 | 0 | 0 | 0 | 0 | 0
  Albumin, Grade 1 | 0 | 0 | 0 | 0 | 0
  Albumin, Grade 2 | 0 | 0 | 0 | 0 | 0
  Albumin, Grade 3 | 0 | 0 | 0 | 0 | 0
  Albumin, Grade 4 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase, Grade 1 | 0 | 0 | 1 | 0 | 0
  Alkaline phosphatase, Grade 2 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase, Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase, Grade 4 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 1 | 1 | 0 | 2 | 1 | 1
  Aspartate aminotransferase, Grade 2 | 1 | 0 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 3 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 4 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Grade 1 | 1 | 1 | 1 | 0 | 0
  Bilirubin, Grade 2 | 0 | 0 | 0 | 0 | 1
  Bilirubin, Grade 3 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Grade 4 | 0 | 0 | 0 | 0 | 0
  Calcium (high), Grade 1 | 0 | 0 | 1 | 1 | 1
  Calcium (high), Grade 2 | 0 | 0 | 0 | 0 | 0
  Calcium (high), Grade 3 | 0 | 0 | 0 | 0 | 0
  Calcium (high), Grade 4 | 0 | 0 | 0 | 0 | 0
  Calcium (low), Grade 1 | 0 | 0 | 0 | 0 | 0
  Calcium (low), Grade 2 | 0 | 0 | 0 | 0 | 0
  Calcium (low), Grade 3 | 0 | 0 | 2 | 0 | 0
  Calcium (low), Grade 4 | 0 | 0 | 0 | 0 | 0
  Creatine kinase, Grade 1 | 0 | 0 | 0 | 1 | 2
  Creatine kinase, Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatine kinase, Grade 3 | 0 | 0 | 0 | 1 | 0
  Creatine kinase, Grade 4 | 2 | 0 | 0 | 0 | 0
  Creatinine, Grade 1 | 0 | 0 | 0 | 0 | 0
  Creatinine, Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatinine, Grade 3 | 1 | 1 | 1 | 0 | 1
  Creatinine, Grade 4 | 0 | 0 | 0 | 0 | 0
  Glucose (high), Grade 1 | 6 | 5 | 10 | 6 | 7
  Glucose (high), Grade 2 | 2 | 0 | 0 | 3 | 3
  Glucose (high), Grade 3 | 0 | 0 | 0 | 1 | 1
  Glucose (high), Grade 4 | 0 | 0 | 0 | 0 | 0
  Glucose (low), Grade 1 | 0 | 0 | 0 | 0 | 1
  Glucose (low), Grade 2 | 1 | 0 | 0 | 0 | 0
  Glucose (low), Grade 3 | 0 | 0 | 0 | 0 | 0
  Glucose (low), Grade 4 | 0 | 0 | 0 | 0 | 0
  Magnesium, Grade 1 | 0 | 0 | 2 | 0 | 0
  Magnesium, Grade 2 | 0 | 0 | 0 | 0 | 0
  Magnesium, Grade 3 | 0 | 0 | 0 | 0 | 0
  Magnesium, Grade 4 | 0 | 0 | 0 | 0 | 0
  Phosphate, Grade 1 | 1 | 1 | 0 | 1 | 4
  Phosphate, Grade 2 | 1 | 1 | 1 | 1 | 0
  Phosphate, Grade 3 | 0 | 0 | 0 | 0 | 0
  Phosphate, Grade 4 | 0 | 0 | 0 | 0 | 0
  Potassium (high), Grade 1 | 0 | 0 | 0 | 0 | 1
  Potassium (high), Grade 2 | 0 | 0 | 0 | 0 | 0
  Potassium (high), Grade 3 | 0 | 0 | 0 | 0 | 0
  Potassium (high), Grade 4 | 0 | 0 | 0 | 0 | 0
  Potassium (low), Grade 1 | 0 | 0 | 2 | 0 | 0
  Potassium (low), Grade 2 | 0 | 0 | 1 | 0 | 0
  Potassium (low), Grade 3 | 0 | 0 | 0 | 0 | 0
  Potassium (low), Grade 4 | 0 | 0 | 0 | 0 | 0
  Sodium (high), Grade 1 | 3 | 0 | 2 | 1 | 5
  Sodium (high), Grade 2 | 0 | 0 | 0 | 0 | 0
  Sodium (high), Grade 3 | 0 | 0 | 0 | 0 | 0
  Sodium (high), Grade 4 | 0 | 0 | 0 | 0 | 0
  Sodium (low), Grade 1 | 0 | 0 | 1 | 0 | 0
  Sodium (low), Grade 2 | 0 | 0 | 0 | 0 | 0
  Sodium (low), Grade 3 | 0 | 0 | 0 | 0 | 0
  Sodium (low), Grade 4 | 0 | 0 | 0 | 0 | 0
  Urate, Grade 1 | 2 | 1 | 1 | 8 | 3
  Urate, Grade 2 | 0 | 0 | 0 | 0 | 0
  Urate, Grade 3 | 0 | 0 | 0 | 0 | 0
  Urate, Grade 4 | 0 | 0 | 0 | 0 | 0
  GFR, Grade 1 | 0 | 0 | 0 | 0 | 0
  GFR, Grade 2 | 0 | 0 | 0 | 0 | 0
  GFR, Grade 3 | 0 | 0 | 0 | 0 | 0
  GFR, Grade 4 | 0 | 0 | 0 | 0 | 0

30. Primary Outcome: Part 2: Number of Participants With Maximum Post-Baseline Grade by Category in Clinical Chemistry Parameters (Up to Day 450-Optional Follow-up)
Description: as for outcome 29
Time Frame: Up to Day 450
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Participants
  Alanine aminotransferase, Grade 1 | 2 | 0 | 3 | 0 | 4
  Alanine aminotransferase, Grade 2 | 0 | 0 | 0 | 1 | 1
  Alanine aminotransferase, Grade 3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase, Grade 4 | 0 | 0 | 0 | 0 | 0
  Albumin, Grade 1 | 0 | 0 | 0 | 0 | 0
  Albumin, Grade 2 | 0 | 0 | 0 | 0 | 0
  Albumin, Grade 3 | 0 | 0 | 0 | 0 | 0
  Albumin, Grade 4 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase, Grade 1 | 0 | 0 | 2 | 0 | 0
  Alkaline phosphatase, Grade 2 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase, Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase, Grade 4 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 1 | 1 | 0 | 2 | 1 | 1
  Aspartate aminotransferase, Grade 2 | 1 | 0 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 3 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase, Grade 4 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Grade 1 | 1 | 1 | 1 | 0 | 0
  Bilirubin, Grade 2 | 0 | 0 | 0 | 0 | 1
  Bilirubin, Grade 3 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Grade 4 | 0 | 0 | 0 | 0 | 0
  Calcium (high), Grade 1 | 0 | 0 | 1 | 1 | 2
  Calcium (high), Grade 2 | 0 | 0 | 0 | 0 | 0
  Calcium (high), Grade 3 | 0 | 0 | 0 | 0 | 0
  Calcium (high), Grade 4 | 0 | 0 | 0 | 0 | 0
  Calcium (low), Grade 1 | 0 | 0 | 0 | 0 | 0
  Calcium (low), Grade 2 | 0 | 0 | 0 | 0 | 0
  Calcium (low), Grade 3 | 0 | 0 | 2 | 0 | 0
  Calcium (low), Grade 4 | 0 | 0 | 0 | 0 | 0
  Creatine kinase, Grade 1 | 0 | 1 | 0 | 2 | 2
  Creatine kinase, Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatine kinase, Grade 3 | 0 | 0 | 0 | 1 | 0
  Creatine kinase, Grade 4 | 2 | 0 | 0 | 0 | 0
  Creatinine, Grade 1 | 0 | 0 | 0 | 0 | 0
  Creatinine, Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatinine, Grade 3 | 1 | 1 | 1 | 0 | 1
  Creatinine, Grade 4 | 0 | 0 | 0 | 0 | 0
  Glucose (high), Grade 1 | 6 | 5 | 11 | 6 | 7
  Glucose (high), Grade 2 | 2 | 0 | 0 | 3 | 3
  Glucose (high), Grade 3 | 0 | 0 | 0 | 1 | 1
  Glucose (high), Grade 4 | 0 | 0 | 0 | 0 | 0
  Glucose (low), Grade 1 | 0 | 0 | 1 | 0 | 1
  Glucose (low), Grade 2 | 1 | 0 | 0 | 0 | 0
  Glucose (low), Grade 3 | 0 | 0 | 0 | 0 | 0
  Glucose (low), Grade 4 | 0 | 0 | 0 | 0 | 0
  Magnesium, Grade 1 | 0 | 0 | 2 | 0 | 0
  Magnesium, Grade 2 | 0 | 0 | 0 | 0 | 0
  Magnesium, Grade 3 | 0 | 0 | 0 | 0 | 0
  Magnesium, Grade 4 | 0 | 0 | 0 | 0 | 0
  Phosphate, Grade 1 | 2 | 1 | 0 | 1 | 4
  Phosphate, Grade 2 | 1 | 1 | 1 | 1 | 0
  Phosphate, Grade 3 | 0 | 0 | 0 | 0 | 0
  Phosphate, Grade 4 | 0 | 0 | 0 | 0 | 0
  Potassium (high), Grade 1 | 0 | 0 | 0 | 0 | 1
  Potassium (high), Grade 2 | 0 | 0 | 0 | 0 | 0
  Potassium (high), Grade 3 | 0 | 0 | 0 | 0 | 0
  Potassium (high), Grade 4 | 0 | 0 | 0 | 0 | 0
  Potassium (low), Grade 1 | 0 | 0 | 2 | 0 | 0
  Potassium (low), Grade 2 | 0 | 0 | 1 | 0 | 0
  Potassium (low), Grade 3 | 0 | 0 | 0 | 0 | 0
  Potassium (low), Grade 4 | 0 | 0 | 0 | 0 | 0
  Sodium (high), Grade 1 | 3 | 0 | 2 | 1 | 6
  Sodium (high), Grade 2 | 0 | 0 | 0 | 0 | 0
  Sodium (high), Grade 3 | 0 | 0 | 0 | 0 | 0
  Sodium (high), Grade 4 | 0 | 0 | 0 | 0 | 0
  Sodium (low), Grade 1 | 0 | 0 | 1 | 0 | 0
  Sodium (low), Grade 2 | 0 | 0 | 0 | 0 | 0
  Sodium (low), Grade 3 | 0 | 0 | 0 | 0 | 0
  Sodium (low), Grade 4 | 0 | 0 | 0 | 0 | 0
  Urate, Grade 1 | 2 | 1 | 2 | 8 | 3
  Urate, Grade 2 | 0 | 0 | 0 | 0 | 0
  Urate, Grade 3 | 0 | 0 | 0 | 0 | 0
  Urate, Grade 4 | 0 | 0 | 0 | 0 | 0
  GFR, Grade 1 | 0 | 0 | 0 | 0 | 0
  GFR, Grade 2 | 0 | 0 | 0 | 0 | 0
  GFR, Grade 3 | 0 | 0 | 0 | 0 | 0
  GFR, Grade 4 | 0 | 0 | 0 | 0 | 0

31. Primary Outcome: Part 1: Change From Baseline in Urine Albumin at Indicated Time Points
Description: Urine samples were collected from participants to assess urine albumin levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Days 8, 30 and Follow-up (Day 60)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Milligram per deciliter
  Day 8 | -0.090 (0.1559) | 0.000 (0.0000) | -0.003 (0.0082)
  Day 30 | -0.090 (0.1559) | 0.000 (0.0000) | -0.003 (0.0082)
  Follow-up (Day 60) | -0.083 (0.1620) | 0.000 (0.0000) | -0.003 (0.0082)

32. Primary Outcome: Part 2: Change From Baseline in Urine Albumin at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 31
Time Frame: Baseline (Day 1 pre-dose), Days 15, 29, 43, 57, 71, 85, 92, 99, 113, 141 and 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
Milligram per deciliter
  Day 15, n=10,6,20,14,14: number analyzed (Participants) | 10 | 6 | 20 | 14 | 14
  Day 15, n=10,6,20,14,14 | 0.484 (1.5305) | 0.000 (0.0000) | 0.004 (0.0157) | -0.044 (0.3593) | 0.054 (2.1129)
  Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, n=10,6,20,13,15 | -0.038 (0.1202) | 0.000 (0.0000) | 0.102 (0.4265) | -0.100 (0.4276) | -0.293 (1.2710)
  Day 43, n=9,6,20,14,15: number analyzed (Participants) | 9 | 6 | 20 | 14 | 15
  Day 43, n=9,6,20,14,15 | -0.076 (0.2267) | 0.027 (0.0653) | 0.047 (0.2247) | 1.356 (5.1498) | -0.263 (1.2876)
  Day 57, n=10,6,20,14,15 | -0.068 (0.2150) | 0.252 (0.6165) | 0.157 (0.6699) | 7.142 (27.1610) | -0.345 (1.2457)
  Day 71, n=10,6,20,14,15 | -0.068 (0.2150) | 0.147 (0.3593) | 0.067 (0.2858) | -0.108 (0.4036) | -0.276 (1.2739)
  Day 85, n=10,6,20,14,15 | -0.068 (0.2150) | 0.260 (0.6369) | 0.105 (0.3408) | -0.028 (0.5206) | -0.249 (1.2805)
  Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 92, n=10,6,19,14,15 | 0.386 (1.4751) | 0.088 (0.1613) | 0.031 (0.1811) | -0.034 (0.1256) | -0.113 (1.6274)
  Day 99, n=10,6,20,14,15 | -0.068 (0.2150) | 0.000 (0.0000) | 0.287 (1.1198) | -0.028 (0.4733) | -0.307 (1.2558)
  Day 113, n=10,6,19,13,15: number analyzed (Participants) | 10 | 6 | 19 | 13 | 15
  Day 113, n=10,6,19,13,15 | -0.020 (0.2766) | 0.057 (0.1388) | 0.376 (1.1353) | -0.060 (0.4801) | -0.342 (1.2507)
  Day 141, n=10,6,20,14,15 | -0.068 (0.2150) | 0.000 (0.0000) | 0.061 (0.2350) | 0.014 (0.3879) | -0.317 (1.2571)
  Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, n=10,6,19,14,15 | -0.068 (0.2150) | 0.223 (0.5471) | 0.436 (1.3939) | -0.095 (0.3555) | -0.317 (1.2678)

33. Primary Outcome: Part 2: Change From Baseline in Urine Albumin at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Urine samples were planned to be collected from participants to evaluate change from Baseline in urine albumin levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was to be calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: Safety Population. Data was not collected for this outcome measure during optional follow-up period.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

34. Primary Outcome: Part 1: Change From Baseline in Urine Creatinine at Indicated Time Points
Description: Urine samples were collected from participants to assess urine creatinine levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Days 8, 30 and Follow-up (Day 60)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Millimoles per liter
  Day 8 | -6.333 (4.8003) | -7.500 (10.8586) | -0.500 (5.4468)
  Day 30 | -4.133 (7.2947) | -7.467 (12.1763) | -0.533 (5.5824)
  Follow-up (Day 60) | 1.800 (14.5000) | -12.500 (12.4386) | -1.917 (6.3031)

35. Primary Outcome: Part 2: Change From Baseline in Urine Creatinine at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 34
Time Frame: Baseline (Day 1 pre-dose), Days 15, 29, 43, 57, 71, 85, 92, 99, 113, 141 and 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
Millimoles per liter
  Day 15, n=10,6,20,14,14: number analyzed (Participants) | 10 | 6 | 20 | 14 | 14
  Day 15, n=10,6,20,14,14 | 1.250 (3.9769) | 3.100 (7.2812) | 1.620 (5.9265) | 0.621 (6.6401) | 1.129 (7.8266)
  Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, n=10,6,20,13,15 | -0.250 (8.1437) | -1.183 (2.2516) | 1.645 (4.2540) | 0.185 (6.7815) | 0.307 (6.2369)
  Day 43, n=9,6,20,14,15: number analyzed (Participants) | 9 | 6 | 20 | 14 | 15
  Day 43, n=9,6,20,14,15 | -1.989 (7.6522) | 1.933 (3.4518) | -0.615 (3.4238) | -1.614 (8.1636) | -0.160 (5.5418)
  Day 57, n=10,6,20,14,15 | 0.730 (6.3381) | 4.283 (6.9975) | -0.005 (4.1111) | -2.336 (7.3438) | -0.707 (5.1370)
  Day 71, n=10,6,20,14,15 | -0.420 (8.0098) | 3.383 (4.1427) | 1.625 (7.4370) | -2.571 (5.5116) | -0.560 (4.8550)
  Day 85, n=10,6,20,14,15 | -0.380 (5.2742) | -0.350 (3.1507) | 1.335 (6.3596) | -1.500 (7.3661) | 0.127 (5.1497)
  Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 92, n=10,6,19,14,15 | 1.900 (6.0566) | 3.367 (4.6224) | 1.353 (5.6700) | -0.679 (8.1936) | -1.013 (5.4487)
  Day 99, n=10,6,20,14,15 | 1.180 (6.5445) | -0.833 (2.7500) | 1.775 (4.6852) | -1.593 (7.3409) | 0.020 (5.1870)
  Day 113, n=10,6,19,13,15: number analyzed (Participants) | 10 | 6 | 19 | 13 | 15
  Day 113, n=10,6,19,13,15 | 1.640 (12.4484) | -0.200 (1.9819) | 0.395 (4.2339) | -0.515 (8.9447) | -1.273 (4.9312)
  Day 141, n=10,6,20,14,15 | -3.440 (8.1759) | -0.150 (4.7218) | 1.090 (4.9374) | 0.464 (7.7548) | -0.713 (5.9545)
  Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, n=10,6,19,14,15 | -1.520 (6.5367) | 2.150 (2.6251) | 2.484 (5.4097) | 0.386 (7.7418) | -2.980 (5.0428)

36. Primary Outcome: Part 2: Change From Baseline in Urine Creatinine at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Urine samples were planned to be collected from participants to evaluate change from Baseline in urine creatinine levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was to be calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: Safety Population. Data was not collected for this outcome measure during optional follow-up period.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

37. Primary Outcome: Part 1: Change From Baseline in Urine Potential of Hydrogen (pH) at Indicated Time Points
Description: Urine samples were collected from participants to assess urine pH levels. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Days 3, 8, 30 and Follow-up (Day 60)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
pH
  Day 3 | 0.333 (0.2887) | 0.167 (0.2887) | 0.083 (0.4916)
  Day 8 | 0.000 (0.0000) | 1.000 (0.5000) | 0.333 (0.6831)
  Day 30 | 0.167 (0.2887) | 0.333 (1.0408) | 0.167 (0.5164)
  Follow-up (Day 60) | 0.167 (0.2887) | 0.500 (1.0000) | 0.250 (0.5244)

38. Primary Outcome: Part 2: Change From Baseline in Urine pH at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 37
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 19 | 14 | 14
pH
  Day 8, n=10,6,19,14,13: number analyzed (Participants) | 10 | 6 | 19 | 14 | 13
  Day 8, n=10,6,19,14,13 | 0.300 (0.9487) | -0.333 (0.8165) | -0.132 (0.7040) | -0.071 (0.4746) | -0.077 (0.6405)
  Day 15, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 15, n=10,6,19,13,14 | 0.200 (0.6325) | -0.500 (1.0488) | -0.026 (0.6341) | -0.154 (0.6887) | 0.000 (0.5547)
  Day 22, n=9,6,19,13,14: number analyzed (Participants) | 9 | 6 | 19 | 13 | 14
  Day 22, n=9,6,19,13,14 | 0.333 (0.7071) | -0.667 (0.5164) | -0.211 (0.7133) | -0.308 (0.6304) | -0.143 (1.0271)
  Day 29, n=10,6,19,12,14: number analyzed (Participants) | 10 | 6 | 19 | 12 | 14
  Day 29, n=10,6,19,12,14 | 0.200 (0.6325) | -0.167 (0.7528) | 0.000 (0.4714) | 0.000 (0.7385) | -0.286 (0.6112)
  Day 36, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 36, n=10,6,19,13,14 | 0.050 (0.8960) | -0.333 (1.0328) | -0.105 (0.4588) | -0.077 (0.6405) | -0.107 (0.7888)
  Day 43, n=9,6,19,13,14: number analyzed (Participants) | 9 | 6 | 19 | 13 | 14
  Day 43, n=9,6,19,13,14 | 0.111 (0.7817) | -0.167 (0.7528) | 0.000 (0.5774) | 0.077 (0.8623) | -0.214 (0.6993)
  Day 50, n=9,6,18,13,14: number analyzed (Participants) | 9 | 6 | 18 | 13 | 14
  Day 50, n=9,6,18,13,14 | 0.000 (0.7071) | -0.167 (1.1690) | 0.000 (0.5941) | -0.231 (0.7250) | 0.036 (0.8872)
  Day 57, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 57, n=10,6,19,13,14 | 0.100 (0.9944) | -0.167 (0.7528) | 0.000 (0.4714) | 0.077 (0.7596) | -0.071 (0.4746)
  Day 64, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 64, n=10,6,19,13,14 | 0.200 (0.6325) | -0.167 (0.7528) | -0.105 (0.6578) | 0.000 (0.5774) | -0.214 (0.5789)
  Day 71, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 71, n=10,6,19,13,14 | 0.200 (0.7888) | -0.167 (0.7528) | 0.000 (0.4714) | 0.077 (0.6405) | -0.071 (0.7300)
  Day 78, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 78, n=10,6,19,13,14 | 0.100 (0.5676) | 0.000 (0.6325) | -0.053 (0.5243) | 0.000 (0.7071) | 0.143 (0.7703)
  Day 85, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 85, n=10,6,19,13,14 | 0.000 (1.0541) | 0.000 (0.8944) | -0.105 (0.6578) | 0.000 (0.5774) | -0.214 (0.5789)
  Day 92, n=10,6,18,13,14: number analyzed (Participants) | 10 | 6 | 18 | 13 | 14
  Day 92, n=10,6,18,13,14 | 0.000 (0.8165) | 0.167 (0.4082) | 0.056 (0.5393) | 0.000 (0.7071) | -0.214 (0.6993)
  Day 99, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 99, n=10,6,19,13,14 | 0.100 (0.5676) | 0.167 (0.9832) | -0.158 (0.5015) | -0.154 (0.9871) | -0.214 (0.5789)
  Day 113, n=10,6,17,12,14: number analyzed (Participants) | 10 | 6 | 17 | 12 | 14
  Day 113, n=10,6,17,12,14 | 0.000 (0.8165) | 0.000 (0.6325) | -0.176 (0.5286) | 0.000 (0.9535) | -0.143 (0.9493)
  Day 141, n=10,6,19,13,14: number analyzed (Participants) | 10 | 6 | 19 | 13 | 14
  Day 141, n=10,6,19,13,14 | 0.300 (0.6749) | 0.167 (0.7528) | 0.053 (0.6213) | -0.077 (0.6405) | -0.143 (0.7703)
  Day 169, n=10,6,18,13,14: number analyzed (Participants) | 10 | 6 | 18 | 13 | 14
  Day 169, n=10,6,18,13,14 | -0.200 (0.7888) | 0.000 (0.6325) | -0.278 (0.4609) | 0.077 (0.6405) | -0.071 (0.4746)

39. Primary Outcome: Part 2: Change From Baseline in Urine pH at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Urine samples were planned to be collected from participants to evaluate change from Baseline in urine pH levels. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was to be calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: Safety Population. Data was not collected for this outcome measure during optional follow-up period.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

40. Primary Outcome: Part 1: Change From Baseline in Urine Specific Gravity at Indicated Time Points
Description: Urine samples were collected from participants to assess urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Days 3, 8, 30 and Follow-up (Day 60)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Ratio
  Day 3 | 0.005 (0.0091) | -0.011 (0.0061) | -0.001 (0.0029)
  Day 8 | 0.003 (0.0081) | -0.014 (0.0151) | 0.000 (0.0087)
  Day 30 | -0.001 (0.0112) | -0.013 (0.0175) | 0.000 (0.0066)
  Follow-up (Day 60) | 0.006 (0.0125) | -0.014 (0.0123) | -0.001 (0.0079)

41. Primary Outcome: Part 2: Change From Baseline in Urine Specific Gravity at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 40
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Ratio
  Day 8, n=10,6,19,15,14: number analyzed (Participants) | 10 | 6 | 19 | 15 | 14
  Day 8, n=10,6,19,15,14 | -0.001 (0.0080) | 0.004 (0.0049) | -0.001 (0.0060) | 0.000 (0.0055) | 0.000 (0.0063)
  Day 15, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 15, n=10,6,20,14,15 | 0.002 (0.0054) | 0.004 (0.0085) | 0.001 (0.0058) | 0.000 (0.0083) | 0.000 (0.0088)
  Day 22, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 22, n=10,6,20,14,15 | -0.001 (0.0082) | 0.003 (0.0045) | -0.001 (0.0073) | 0.001 (0.0063) | 0.000 (0.0070)
  Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, n=10,6,20,13,15 | 0.001 (0.0098) | -0.001 (0.0060) | 0.001 (0.0052) | 0.000 (0.0051) | 0.001 (0.0064)
  Day 36, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 36, n=10,6,20,14,15 | 0.004 (0.0100) | 0.002 (0.0067) | -0.002 (0.0065) | -0.001 (0.0067) | -0.003 (0.0082)
  Day 43, n=9,6,20,14,15: number analyzed (Participants) | 9 | 6 | 20 | 14 | 15
  Day 43, n=9,6,20,14,15 | -0.003 (0.0098) | 0.002 (0.0060) | 0.000 (0.0050) | -0.001 (0.0070) | 0.000 (0.0064)
  Day 50, n=9,6,19,14,15: number analyzed (Participants) | 9 | 6 | 19 | 14 | 15
  Day 50, n=9,6,19,14,15 | -0.003 (0.0081) | 0.002 (0.0079) | -0.002 (0.0065) | -0.001 (0.0095) | 0.000 (0.0076)
  Day 57, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 57, n=10,6,20,14,15 | 0.000 (0.0082) | 0.005 (0.0078) | -0.001 (0.0044) | -0.003 (0.0073) | 0.000 (0.0069)
  Day 64, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 64, n=10,6,20,14,15 | -0.002 (0.0103) | 0.003 (0.0093) | 0.000 (0.0055) | -0.001 (0.0059) | 0.001 (0.0052)
  Day 71, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 71, n=10,6,20,14,15 | -0.001 (0.0100) | 0.003 (0.0052) | 0.001 (0.0072) | -0.003 (0.0059) | 0.001 (0.0053)
  Day 78, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 78, n=10,6,20,14,15 | -0.002 (0.0069) | 0.002 (0.0022) | 0.000 (0.0078) | -0.004 (0.0085) | -0.001 (0.0081)
  Day 85, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 85, n=10,6,20,14,15 | 0.001 (0.0074) | -0.002 (0.0023) | 0.000 (0.0057) | -0.003 (0.0074) | 0.000 (0.0058)
  Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 92, n=10,6,19,14,15 | 0.001 (0.0070) | 0.002 (0.0051) | 0.001 (0.0063) | -0.002 (0.0079) | 0.000 (0.0058)
  Day 99, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 99, n=10,6,20,14,15 | 0.002 (0.0081) | -0.001 (0.0039) | 0.001 (0.0050) | -0.002 (0.0061) | 0.000 (0.0048)
  Day 113, n=10,6,18,13,15: number analyzed (Participants) | 10 | 6 | 18 | 13 | 15
  Day 113, n=10,6,18,13,15 | 0.000 (0.0101) | 0.000 (0.0043) | 0.000 (0.0054) | -0.001 (0.0090) | -0.001 (0.0047)
  Day 141, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 141, n=10,6,20,14,15 | -0.003 (0.0107) | -0.001 (0.0068) | 0.001 (0.0056) | 0.000 (0.0086) | 0.000 (0.0066)
  Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, n=10,6,19,14,15 | -0.001 (0.0072) | 0.002 (0.0053) | 0.001 (0.0047) | 0.000 (0.0077) | -0.003 (0.0052)

42. Primary Outcome: Part 2: Change From Baseline in Urine Specific Gravity at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Urine samples were planned to be collected from participants to evaluate change from Baseline in urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was to be calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: Safety Population. Data was not collected for this outcome measure during optional follow-up period.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

43. Primary Outcome: Part 1: Change From Baseline in Urobilinogen at Indicated Time Points
Description: Urine samples were collected from participants to assess urobilinogen levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Days 3, 8, 30 and Follow-up (Day 60)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Milligram per deciliter
  Day 3 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 8 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 30 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Follow-up (Day 60) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)

44. Primary Outcome: Part 2: Change From Baseline in Urobilinogen at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 43
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Milligram per deciliter
  Day 8, n=10,6,19,15,14: number analyzed (Participants) | 10 | 6 | 19 | 15 | 14
  Day 8, n=10,6,19,15,14 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 15, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 15, n=10,6,20,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.090 (0.4025) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 22, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 22, n=10,6,20,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, n=10,6,20,13,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.120 (0.4648)
  Day 36, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 36, n=10,6,20,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.120 (0.4648)
  Day 43, n=9,6,20,14,15: number analyzed (Participants) | 9 | 6 | 20 | 14 | 15
  Day 43, n=9,6,20,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.180 (0.5540) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 50, n=9,6,19,14,15: number analyzed (Participants) | 9 | 6 | 19 | 14 | 15
  Day 50, n=9,6,19,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 57, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 57, n=10,6,20,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.090 (0.4025) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 64, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 64, n=10,6,20,14,15 | 0.180 (0.5692) | 0.000 (0.0000) | 0.180 (0.5540) | 0.000 (0.0000) | 0.240 (0.6334)
  Day 71, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 71, n=10,6,19,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.240 (0.6334)
  Day 78, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 78, n=10,6,20,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.180 (0.5540) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 85, n=10,6,20,14,14: number analyzed (Participants) | 10 | 6 | 20 | 14 | 14
  Day 85, n=10,6,20,14,14 | 0.000 (0.0000) | 0.000 (0.0000) | 0.090 (0.4025) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 92, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 92, n=10,6,19,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.189 (0.5675) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 99, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 99, n=10,6,19,14,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.120 (0.4648)
  Day 113, n=10,6,17,13,15: number analyzed (Participants) | 10 | 6 | 17 | 13 | 15
  Day 113, n=10,6,17,13,15 | 0.000 (0.0000) | 0.000 (0.0000) | 0.106 (0.4366) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 141, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 141, n=10,6,19,14,15 | 0.180 (0.5692) | 0.000 (0.0000) | 0.095 (0.4129) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 169, n=10,6,19,14,14: number analyzed (Participants) | 10 | 6 | 19 | 14 | 14
  Day 169, n=10,6,19,14,14 | 0.000 (0.0000) | 0.000 (0.0000) | 0.095 (0.4129) | 0.000 (0.0000) | 0.129 (0.4811)

45. Primary Outcome: Part 2: Change From Baseline in Urobilinogen at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Urine samples were planned to be collected from participants to evaluate change from Baseline in urobilinogen. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Change from Baseline was to be calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: Safety Population. Data was not collected for this outcome measure during optional follow-up period.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

46. Primary Outcome: Part 1: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Electrocardiograms were obtained after 5 minutes of rest in the semi-supine or supine position using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings have been presented. Clinical significance was based on the medical and scientific judgement of the investigator or qualified designee.
Time Frame: Day 1: 2 hours, Day 1: 4 hours, Day 1: 8 hours, Day 3, Day 8 and Day 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants
  Abnormal NCS, Day 1: 2 hour, n=3,3,6 | 2 | 1 | 5
  Abnormal CS, Day 1: 2 hour, n=3,3,6 | 0 | 0 | 0
  Abnormal NCS, Day 1: 4 hour, n=3,3,6 | 2 | 2 | 3
  Abnormal CS, Day 1: 4 hour, n=3,3,6 | 0 | 0 | 0
  Abnormal NCS, Day 1: 8 hour, n=3,3,6 | 2 | 2 | 5
  Abnormal CS, Day 1: 8 hour, n=3,3,6 | 0 | 0 | 0
  Abnormal NCS, Day 3, n=3,3,6 | 2 | 1 | 3
  Abnormal CS, Day 3, n=3,3,6 | 0 | 0 | 0
  Abnormal NCS, Day 8, n=2,3,6: number analyzed (Participants) | 2 | 3 | 6
  Abnormal NCS, Day 8, n=2,3,6 | 1 | 1 | 2
  Abnormal CS, Day 8, n=2,3,6: number analyzed (Participants) | 2 | 3 | 6
  Abnormal CS, Day 8, n=2,3,6 | 0 | 0 | 0
  Abnormal NCS, Day 30, n=3,3,6 | 2 | 1 | 2
  Abnormal CS, Day 30, n=3,3,6 | 0 | 0 | 0

47. Primary Outcome: Part 2: Number of Participants With Abnormal ECG Findings (Up to Day 169-Interim Analysis)
Description: Electrocardiogram were obtained after 5 minutes of rest in the semi-supine or supine position using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals. CS and NCS abnormal ECG findings have been presented. Clinical significance was based on the medical and scientific judgement of the investigator or qualified designee.
Time Frame: Days 29, 57, 85 and 169
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
Participants
  Day 29, NCS, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, NCS, n=10,6,20,13,15 | 2 | 2 | 6 | 6 | 5
  Day 29, CS, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, CS, n=10,6,20,13,15 | 0 | 0 | 0 | 0 | 0
  Day 57, NCS, n=10,6,20,14,15 | 5 | 3 | 6 | 3 | 6
  Day 57, CS, n=10,6,20,14,15 | 0 | 0 | 0 | 0 | 0
  Day 85, NCS, n=10,6,20,14,15 | 3 | 3 | 4 | 4 | 4
  Day 85, CS, n=10,6,20,14,15 | 0 | 0 | 0 | 0 | 0
  Day 169, NCS, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, NCS, n=10,6,19,14,15 | 2 | 2 | 4 | 5 | 5
  Day 169, CS, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, CS, n=10,6,19,14,15 | 0 | 0 | 0 | 0 | 0

48. Primary Outcome: Part 2: Number of Participants With Abnormal ECG Findings (Up to Day 450-Optional Follow-up)
Description: ECGs were planned to be obtained after 5 minutes of rest in the semi-supine or supine position using ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTcF intervals.
Time Frame: Days 270, 360 and 450
Population: Safety Population. Data was not collected for this outcome measure during optional follow-up period.
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

49. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment were categorized as SAE.
Time Frame: Up to Day 60
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants
  AEs | 1 | 0 | 1
  SAEs | 0 | 0 | 0

50. Primary Outcome: Part 2: Number of Participants With AEs and SAEs (Up to Day 169-Interim Analysis)
Description: as for outcome 49
Time Frame: Up to Day 169
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Participants
  AEs | 9 | 4 | 16 | 11 | 12
  SAEs | 1 | 0 | 0 | 2 | 0

51. Primary Outcome: Part 2: Number of Participants With AEs and SAEs (Up to Day 450-Optional Follow-up)
Description: as for outcome 49
Time Frame: Up to Day 450
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Participants
  AEs | 9 | 4 | 18 | 11 | 12
  SAEs | 1 | 0 | 0 | 2 | 1

52. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to the Time of the Last Quantifiable Concentration (AUC[0-t]) for GSK3389404
Description: Blood samples were collected to measure AUC(0-t) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population comprised of all participants in the Safety population for whom at least one evaluable pharmacokinetic sample were obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 6
Hours*nanogram per milliliter | 1230 (14.3) | 17000 (39.5)

53. Primary Outcome: Part 2: AUC (0-t) for GSK3389404
Description: as for outcome 52
Time Frame: Day 1 (Pre-dose and at 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose), Days 29 and 57 (Pre-dose and at 1, 2, 3 hours post-dose), Day 169
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 6 | 6 | 3 | 3
Hours*nanogram per milliliter | 1930 (21.4) | 5920 (36.2) | 12000 (38.5) | 14400 (49.1)

54. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-infinity]) for GSK3389404
Description: Blood samples were collected to measure AUC (0-infinity) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 2 | 3
Hours*nanogram per milliliter | 1460 (15.5) | 17100 (23.2)

55. Primary Outcome: Part 2: AUC (0-infinity) for GSK3389404
Description: as for outcome 54
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 6 | 6 | 3 | 3
Hours*nanogram per milliliter | 2030 (17.7) | 5990 (35.3) | 12300 (37.5) | 14600 (47.3)

56. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of GSK3389404
Description: Blood samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 6
Nanogram per milliliter | 227 (11.0) | 1880 (72.4)

57. Primary Outcome: Part 2: Cmax of GSK3389404
Description: as for outcome 56
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 6 | 6 | 3 | 3
Nanogram per milliliter | 214 (54.3) | 865 (41.3) | 1660 (34.4) | 1940 (78.2)

58. Primary Outcome: Part 1: Time to Achieve Cmax (Tmax) of GSK3389404
Description: Blood samples were collected to measure Tmax at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 6
Hours | 1.40 [1.33 to 2.00] | 3.50 [1.93 to 6.00]

59. Primary Outcome: Part 2: Tmax of GSK3389404
Description: as for outcome 58
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 6 | 6 | 3 | 3
Hours | 2.04 [0.90 to 3.98] | 3.46 [1.98 to 5.98] | 4.05 [2.02 to 6.03] | 4.02 [2.98 to 4.07]

60. Primary Outcome: Part 1: Apparent Terminal Phase Half-life(t1/2) of GSK3389404
Description: Blood samples were collected to measure t1/2 at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 2 | 3
Hours | 3.12 (54.7) | 4.31 (3.7)

61. Primary Outcome: Part 2: t1/2 of GSK3389404
Description: as for outcome 60
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 6 | 6 | 3 | 3
Hours | 3.90 (55.0) | 3.24 (26.0) | 4.24 (29.5) | 2.89 (48.4)

62. Primary Outcome: Part 1: Apparent Subcutaneous Plasma Clearance (CL/F) of GSK3389404
Description: Blood samples were collected to measure CL/F at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per hour
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 2 | 3
Liters per hour | 20.6 [-7.914 to 49.34] | 7.03 [3.090 to 11.22]

63. Primary Outcome: Part 2: CL/F of GSK3389404
Description: as for outcome 62
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per hour
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 6 | 6 | 3 | 3
Liters per hour | 14.8 [12.37 to 17.57] | 10.0 [6.960 to 14.03] | 9.75 [1.914 to 18.41] | 8.23 [0.02305 to 17.51]

64. Primary Outcome: Part 1: Number of Participants Achieving Response Rate (RR) Based on Reduction of Hepatitis B Surface Antigen (HBsAg) Level From Baseline
Description: The RR was based on the proportion of participants with at least a 1.5 logarithm to the base 10 (log10) international units per milliliter (IU/mL) reduction of HBsAg levels from Baseline at any time up to Day 60. Number of participants who achieved >1.5 log10 IU/mL decrease in HBsAg levels at any time up to Day 60 are presented.
Time Frame: Up to Day 60
Population: Intent-To-Treat (ITT) Population comprised of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

65. Primary Outcome: Part 2: Number of Participants Achieving RR Based on Reduction of HBsAg Level From Baseline
Description: The RR was based on the proportion of participants with at least a 1.5 log10 IU/mL reduction of HBsAg levels from Baseline at any time up to Day 85. Number of participants who achieved >1.5 log10 IU/mL decrease in HBsAg levels at any time up to Day 85 are presented.
Time Frame: Up to Day 85
Population: ITT Population. Data is presented only for interim analysis; since this analysis was not planned for optional follow-up period (up to Day 450).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Participants | 0 | 0 | 1 | 1 | 1

66. Secondary Outcome: Part 1: Change From Baseline in log10 Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Viral Load in Plasma at Indicated Time Points
Description: Blood samples were collected from participants to assess HBV DNA viral load. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Log10 change from Baseline was calculated as log10(Post-Dose Visit Value/Baseline).
Time Frame: Baseline (Day 1 pre-dose), Day 1: 8 hours, Days 3, 8, 15, 22, 30 and 60
Population: Pharmacodynamic Population comprised of all participants in the Safety Population who provided evaluable pharmacodynamic data. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 2 | 3 | 6
Log10 (IU/mL)
  Day 1: 8 hour, n=2,3,5: number analyzed (Participants) | 2 | 3 | 5
  Day 1: 8 hour, n=2,3,5 | -0.19 (0.202) | -0.03 (0.055) | 0.50 (0.716)
  Day 3, n=2,3,6 | -0.06 (0.065) | 0.41 (0.754) | 0.20 (0.539)
  Day 8, n=2,3,6 | 0.06 (0.265) | 0.37 (0.788) | -0.02 (0.075)
  Day 15, n=2,3,6 | 0.17 (0.173) | -0.05 (0.086) | -0.17 (0.317)
  Day 22, n=2,3,6 | 0.16 (0.224) | -0.07 (0.114) | -0.09 (0.165)
  Day 30, n=2,3,6 | -0.12 (0.077) | 0.34 (0.821) | 0.13 (0.573)
  Day 60, n=2,3,6 | -0.30 (0.292) | -0.04 (0.075) | 0.12 (0.199)

67. Secondary Outcome: Part 2: Change From Baseline in log10 HBV DNA Viral Load in Plasma at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 66
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 169
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Log10 (IU/mL) | -0.128 (0.4044) | -0.426 (0.6603) | -0.643 (0.6594) | -0.341 (0.7591) | -0.256 (0.5295)

68. Secondary Outcome: Part 2: Change From Baseline in log10 HBV DNA Viral Load in Plasma at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: as for outcome 66
Time Frame: Baseline (Day 1 pre-dose) and Up to Day 450
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Log10 (IU/mL) | -0.128 (0.4044) | -0.426 (0.6603) | -0.643 (0.6594) | -0.426 (0.7893) | -0.256 (0.5295)

69. Secondary Outcome: Part 1: Change From Baseline in log10 Hepatitis B Virus Surface Antigen (HBsAg) Levels in Plasma at Indicated Time Points
Description: Blood samples were collected from participants to assess HBsAg levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Log10 change from Baseline was calculated as log10(Post-Dose Visit Value/Baseline).
Time Frame: Baseline (Day 1 pre-dose) and Day 1: 8 hours, Days 3, 8, 15, 22, 30 and 60
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 6
Log10 (IU/mL)
  Day 1: 8 hour | -0.03 (0.027) | 0.02 (0.023) | -0.02 (0.032)
  Day 3 | 0.01 (0.016) | 0.00 (0.014) | -0.05 (0.038)
  Day 8 | -0.01 (0.078) | 0.01 (0.051) | -0.09 (0.079)
  Day 15 | 0.00 (0.066) | -0.02 (0.043) | -0.10 (0.075)
  Day 22 | 0.03 (0.052) | -0.04 (0.066) | -0.14 (0.114)
  Day 30 | -0.01 (0.038) | -0.02 (0.021) | -0.12 (0.139)
  Day 60 | -0.00 (0.064) | 0.01 (0.057) | -0.05 (0.038)

70. Secondary Outcome: Part 2: Change From Baseline in log10 HBsAg Levels in Plasma at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 69
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: ITT Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 6 | 20 | 15 | 15
Log10 (IU/mL)
  Day 8, n=10,6,20,15,15 | -0.0149 (0.07545) | -0.0057 (0.05207) | -0.0376 (0.08685) | -0.0573 (0.03889) | -0.0944 (0.08417)
  Day 15, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 15, n=10,6,20,14,15 | -0.0175 (0.07296) | -0.0296 (0.03871) | -0.0872 (0.12991) | -0.0690 (0.06427) | -0.2103 (0.13356)
  Day 22, n=10,6,20,15,15 | -0.0248 (0.06304) | -0.0302 (0.03943) | -0.1543 (0.16457) | -0.1200 (0.09169) | -0.3345 (0.17978)
  Day 29, n=10,6,20,13,15: number analyzed (Participants) | 10 | 6 | 20 | 13 | 15
  Day 29, n=10,6,20,13,15 | -0.0252 (0.06330) | -0.0416 (0.07503) | -0.2197 (0.25896) | -0.1793 (0.08003) | -0.4512 (0.22095)
  Day 36, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 36, n=10,6,20,14,15 | -0.0280 (0.06764) | -0.0895 (0.06557) | -0.2650 (0.28541) | -0.2105 (0.08617) | -0.4798 (0.21487)
  Day 43, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 43, n=10,6,20,14,15 | -0.0334 (0.08425) | -0.1010 (0.06003) | -0.2671 (0.31301) | -0.2370 (0.12134) | -0.4923 (0.23961)
  Day 50, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 50, n=10,6,19,14,15 | -0.0118 (0.06170) | -0.0959 (0.06731) | -0.3131 (0.28058) | -0.2603 (0.10027) | -0.5600 (0.31750)
  Day 57, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 57, n=10,6,20,14,15 | -0.0307 (0.05677) | -0.1250 (0.08371) | -0.3171 (0.27547) | -0.2925 (0.09666) | -0.5962 (0.34848)
  Day 64, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 64, n=10,6,20,14,15 | -0.0178 (0.07303) | -0.1388 (0.08620) | -0.3307 (0.25414) | -0.3628 (0.20369) | -0.6261 (0.40132)
  Day 71, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 71, n=10,6,20,14,15 | -0.0124 (0.06586) | -0.1689 (0.13050) | -0.3249 (0.24978) | -0.3722 (0.28298) | -0.6357 (0.42715)
  Day 78, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 78, n=10,6,19,14,15 | -0.0130 (0.08312) | -0.1065 (0.09399) | -0.3438 (0.29089) | -0.4532 (0.46786) | -0.7088 (0.57034)
  Day 85, n=9,6,20,14,14: number analyzed (Participants) | 9 | 6 | 20 | 14 | 14
  Day 85, n=9,6,20,14,14 | -0.0212 (0.08048) | -0.1312 (0.06855) | -0.3374 (0.31804) | -0.4429 (0.50368) | -0.7531 (0.64776)
  Day 92, n=10,6,19,14,13: number analyzed (Participants) | 10 | 6 | 19 | 14 | 13
  Day 92, n=10,6,19,14,13 | -0.0462 (0.12954) | -0.1431 (0.08963) | -0.3411 (0.22578) | -0.4291 (0.56931) | -0.6794 (0.62942)
  Day 99, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 99, n=10,6,20,14,15 | -0.0502 (0.10885) | -0.1084 (0.06213) | -0.3018 (0.20862) | -0.4327 (0.55294) | -0.5981 (0.48977)
  Day 113, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 113, n=10,6,20,14,15 | -0.0395 (0.08067) | -0.0874 (0.05607) | -0.2389 (0.12015) | -0.3612 (0.55395) | -0.4228 (0.36072)
  Day 141, n=10,6,20,14,15: number analyzed (Participants) | 10 | 6 | 20 | 14 | 15
  Day 141, n=10,6,20,14,15 | -0.0132 (0.09127) | -0.0417 (0.04609) | -0.1420 (0.10442) | -0.2246 (0.38875) | -0.2729 (0.23994)
  Day 169, n=10,6,19,14,15: number analyzed (Participants) | 10 | 6 | 19 | 14 | 15
  Day 169, n=10,6,19,14,15 | -0.0046 (0.09142) | -0.0295 (0.03644) | -0.0975 (0.08478) | -0.1038 (0.22824) | -0.1822 (0.21674)

71. Secondary Outcome: Part 2: Change From Baseline in log10 HBsAg Level in Plasma at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: Blood samples were collected from participants to assess HBsAg level. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Log10 change from Baseline was calculated as log10(Post-Dose Visit Value/Baseline).
Time Frame: Baseline (Day 1 pre-dose), Day 270, Day 360 and Day 450
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 10 | 5 | 17 | 13 | 15
Log10 (IU/mL)
  Day 270, n=10,5,17,13,15 | -0.0177 (0.08736) | 0.0308 (0.07338) | 0.0627 (0.21462) | 0.0400 (0.05783) | -0.0047 (0.35902)
  Day 360, n=10,5,17,12,14: number analyzed (Participants) | 10 | 5 | 17 | 12 | 14
  Day 360, n=10,5,17,12,14 | -0.0723 (0.11352) | -0.0397 (0.06918) | -0.0265 (0.08988) | -0.0239 (0.07252) | -0.1175 (0.21454)
  Day 450, n=9,5,17,11,15: number analyzed (Participants) | 9 | 5 | 17 | 11 | 15
  Day 450, n=9,5,17,11,15 | -0.1282 (0.09933) | -0.0551 (0.11173) | -0.0615 (0.08487) | -0.0350 (0.08041) | -0.1557 (0.18720)

72. Secondary Outcome: Part 1: Change From Baseline in log10 Hepatitis B Virus E-antigen (HBeAg) Levels in Plasma at Indicated Time Points
Description: Blood samples were collected from participants to assess HBeAg levels. Baseline was defined as the last assessment before the first dose of the study treatment (Day 1 pre-dose). Log10 change from Baseline was calculated as log10(Post-Dose Visit Value/Baseline).
Time Frame: Baseline (Day 1 pre-dose) and Day 1: 8 hours, Days 3, 8, 15, 22, 30 and 60
Population: Pharmacodynamic Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 3 | 5
Log10 (IU/mL)
  Day 1: 8 hour, n=3,3,5 | 0.15 (0.237) | -0.03 (0.053) | 0.00 (0.000)
  Day 3, n=3,3,4: number analyzed (Participants) | 3 | 3 | 4
  Day 3, n=3,3,4 | -0.01 (0.020) | -0.02 (0.039) | 0.00 (0.000)
  Day 8, n=3,3,4: number analyzed (Participants) | 3 | 3 | 4
  Day 8, n=3,3,4 | 0.02 (0.036) | 0.03 (0.044) | 0.94 (1.885)
  Day 15, n=3,3,4: number analyzed (Participants) | 3 | 3 | 4
  Day 15, n=3,3,4 | 0.02 (0.036) | -0.01 (0.025) | 0.00 (0.000)
  Day 22, n=3,3,4: number analyzed (Participants) | 3 | 3 | 4
  Day 22, n=3,3,4 | 0.03 (0.052) | 0.01 (0.012) | 0.08 (0.151)
  Day 30, n=3,3,4: number analyzed (Participants) | 3 | 3 | 4
  Day 30, n=3,3,4 | 0.22 (0.331) | -0.02 (0.039) | 0.17 (0.342)
  Day 60, n=3,3,4: number analyzed (Participants) | 3 | 3 | 4
  Day 60, n=3,3,4 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

73. Secondary Outcome: Part 2: Change From Baseline in log10 HBeAg Levels in Plasma at Indicated Time Points (Up to Day 169-Interim Analysis)
Description: as for outcome 72
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, 113, 141 and 169
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 7 | 6 | 15 | 11 | 10
Log10 (IU/mL)
  Day 8, n=7,6,15,11,10 | 0.039 (0.0750) | 0.023 (0.0565) | 0.010 (0.0555) | -0.051 (0.0802) | 0.012 (0.0586)
  Day 15, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 15, n=7,6,13,10,9 | 0.101 (0.2223) | -0.030 (0.0516) | -0.020 (0.0519) | -0.044 (0.0728) | -0.009 (0.0976)
  Day 22, n=7,6,13,11,9: number analyzed (Participants) | 7 | 6 | 13 | 11 | 9
  Day 22, n=7,6,13,11,9 | 0.008 (0.0215) | -0.008 (0.0203) | -0.054 (0.0732) | -0.068 (0.1008) | -0.081 (0.1414)
  Day 29, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 29, n=7,6,13,10,9 | 0.050 (0.0937) | 0.003 (0.0552) | -0.049 (0.1086) | -0.059 (0.0959) | -0.039 (0.2732)
  Day 36, n=7,6,12,10,9: number analyzed (Participants) | 7 | 6 | 12 | 10 | 9
  Day 36, n=7,6,12,10,9 | 0.120 (0.2791) | -0.028 (0.0695) | -0.129 (0.2040) | -0.062 (0.1232) | -0.057 (0.1380)
  Day 43, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 43, n=7,6,13,10,9 | 0.008 (0.0397) | -0.006 (0.0603) | -0.113 (0.1285) | -0.067 (0.1146) | 0.013 (0.5325)
  Day 50, n=7,6,12,10,9: number analyzed (Participants) | 7 | 6 | 12 | 10 | 9
  Day 50, n=7,6,12,10,9 | 0.007 (0.0186) | -0.012 (0.0574) | -0.091 (0.1283) | 0.017 (0.3365) | -0.122 (0.1563)
  Day 57, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 57, n=7,6,13,10,9 | 0.002 (0.0111) | -0.024 (0.0592) | -0.110 (0.1288) | -0.040 (0.1506) | -0.068 (0.2413)
  Day 64, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 64, n=7,6,13,10,9 | 0.008 (0.0139) | 0.018 (0.1297) | -0.120 (0.1296) | -0.073 (0.1216) | -0.109 (0.1562)
  Day 71, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 71, n=7,6,13,10,9 | 0.061 (0.1113) | 0.001 (0.0457) | -0.111 (0.1141) | -0.060 (0.1002) | -0.101 (0.1618)
  Day 78, n=7,6,12,10,9: number analyzed (Participants) | 7 | 6 | 12 | 10 | 9
  Day 78, n=7,6,12,10,9 | -0.027 (0.1334) | 0.086 (0.2363) | -0.100 (0.1224) | -0.071 (0.1232) | -0.118 (0.1636)
  Day 85, n=6,6,13,10,8: number analyzed (Participants) | 6 | 6 | 13 | 10 | 8
  Day 85, n=6,6,13,10,8 | 0.018 (0.0438) | 0.059 (0.1518) | -0.101 (0.1161) | -0.017 (0.1918) | -0.117 (0.1544)
  Day 92, n=7,6,12,10,9: number analyzed (Participants) | 7 | 6 | 12 | 10 | 9
  Day 92, n=7,6,12,10,9 | -0.019 (0.1253) | -0.004 (0.0551) | -0.089 (0.0944) | -0.042 (0.0926) | -0.085 (0.1200)
  Day 99, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 99, n=7,6,13,10,9 | -0.025 (0.1243) | 0.010 (0.0624) | -0.080 (0.0946) | -0.002 (0.1413) | -0.085 (0.1189)
  Day 113, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 113, n=7,6,13,10,9 | 0.015 (0.0628) | -0.003 (0.0666) | -0.040 (0.0773) | -0.022 (0.0543) | -0.011 (0.1237)
  Day 141, n=7,6,13,10,9: number analyzed (Participants) | 7 | 6 | 13 | 10 | 9
  Day 141, n=7,6,13,10,9 | 0.209 (0.4253) | 0.017 (0.1427) | -0.040 (0.1006) | -0.020 (0.0405) | 0.015 (0.0858)
  Day 169, n=7,6,12,9,9: number analyzed (Participants) | 7 | 6 | 12 | 9 | 9
  Day 169, n=7,6,12,9,9 | 0.093 (0.1966) | 0.004 (0.0398) | -0.099 (0.2382) | -0.028 (0.0556) | 0.022 (0.0883)

74. Secondary Outcome: Part 2: Change From Baseline in log10 HBeAg Level in Plasma at Indicated Time Points (Up to Day 450-Optional Follow-up)
Description: as for outcome 72
Time Frame: Baseline (Day 1 pre-dose), Day 270, Day 360 and Day 450
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 7 | 5 | 12 | 10 | 9
Log10 (IU/mL)
  Day 270, n=7,5,11,10,9: number analyzed (Participants) | 7 | 5 | 11 | 10 | 9
  Day 270, n=7,5,11,10,9 | 0.050 (0.1771) | -0.028 (0.3263) | -0.120 (0.3325) | -0.041 (0.0670) | 0.014 (0.0877)
  Day 360, n=7,5,11,9,9: number analyzed (Participants) | 7 | 5 | 11 | 9 | 9
  Day 360, n=7,5,11,9,9 | -0.153 (0.3744) | -0.122 (0.2189) | -0.084 (0.2531) | -0.035 (0.0689) | -0.003 (0.1408)
  Day 450, n=6,5,12,8,9: number analyzed (Participants) | 6 | 5 | 12 | 8 | 9
  Day 450, n=6,5,12,8,9 | 0.000 (0.0000) | -0.119 (0.1866) | -0.088 (0.2225) | -0.155 (0.2663) | -0.035 (0.0627)

75. Secondary Outcome: Part 1: AUC(0-t) for Metabolite of GSK3389404 (ISIS 505358)
Description: as for outcome 52
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 3 | 6
Hours*nanogram per milliliter | NA (NA) — NA indicates that the data is not available since data is below limit of quantification. | 44.2 (419.1)

76. Secondary Outcome: Part 2: AUC(0-t) for Metabolite of GSK3389404 (ISIS 505358)
Description: as for outcome 52
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 1 | 1 | 3
Hours*nanogram per milliliter |  | NA (NA) — NA indicates that the data is not available since data is below limit of quantification. | NA (NA) — NA indicates that the data is not available since data is below limit of quantification. | 17.1 (169.7)

77. Secondary Outcome: Part 1: Cmax of GSK3389404 Metabolite (ISIS 505358)
Description: as for outcome 56
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 5
Nanogram per milliliter |  | 2.93 (60.1)

78. Secondary Outcome: Part 2: Cmax of GSK3389404 Metabolite (ISIS 505358)
Description: as for outcome 56
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 1 | 1 | 3
Nanogram per milliliter |  | NA (NA) — NA indicates that the data is not available since data is below limit of quantification. | NA (NA) — NA indicates that the data is not available since data is below limit of quantification. | 2.91 (77.5)

79. Secondary Outcome: Part 1: Tmax of GSK3389404 Metabolite (ISIS 505358)
Description: as for outcome 58
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 5
Hours |  | 7.88 [4.00 to 48.08]

80. Secondary Outcome: Part 2: Tmax of GSK3389404 Metabolite (ISIS 505358)
Description: as for outcome 58
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 1 | 1 | 3
Hours |  | 7.93 [7.93 to 7.93] | 7.93 [7.93 to 7.93] | 8.00 [4.05 to 8.02]

81. Secondary Outcome: Part 1: t1/2 of GSK3389404 Metabolite (ISIS 505358)
Description: as for outcome 60
Time Frame: Day 1 (Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose), Days 3, 8 and 30
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 1
Hours |  | 18.75 (NA) — NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.

82. Secondary Outcome: Part 2: t1/2 of GSK3389404 Metabolite (ISIS 505358)
Description: as for outcome 60
Time Frame: as for outcome 53
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 1
Hours |  |  |  | 10.66 (NA) — NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.

ADVERSE EVENTS:
Time Frame: SAEs and non-SAEs were collected from the start of study treatment up to Day 60 for Part 1 and up to Day 450 (inclusion of optional follow-up duration) for Part 2
Description: SAEs and AEs were reported treatment-wise for the Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment. No participants were enrolled in Part 1 GSK3389404 60 mg and 240 mg arm groups hence no SAEs and AEs were reported for these two groups.
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 120 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg Weekly | Part 2: GSK3389404 60 mg Weekly | Part 2: GSK3389404 120 mg Bi-weekly | Part 2: GSK3389404 120 mg Weekly
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/10 | 0/6 | 0/20 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 1/10 | 0/6 | 0/20 | 2/15 | 1/15
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/6 | 9/10 | 4/6 | 18/20 | 11/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=3) | Part 1: GSK3389404 30 mg (N=3) | Part 1: GSK3389404 120 mg (N=6) | Part 2: Placebo (N=10) | Part 2: GSK3389404 30 mg Weekly (N=6) | Part 2: GSK3389404 60 mg Weekly (N=20) | Part 2: GSK3389404 120 mg Bi-weekly (N=15) | Part 2: GSK3389404 120 mg Weekly (N=15)
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Putamen haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=3) | Part 1: GSK3389404 30 mg (N=3) | Part 1: GSK3389404 120 mg (N=6) | Part 2: Placebo (N=10) | Part 2: GSK3389404 30 mg Weekly (N=6) | Part 2: GSK3389404 60 mg Weekly (N=20) | Part 2: GSK3389404 120 mg Bi-weekly (N=15) | Part 2: GSK3389404 120 mg Weekly (N=15)
Malaise (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 6 | 2 | 2
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Systemic viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Urine albumin/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Complement factor C3 decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Reticulocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Borderline glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mumps (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT03020745/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT03020745/SAP_002.pdf